

### Statistical Analysis Plan

# Zealand Pharma A/S

### ZP4207-21052

A Phase 3, single-administration open-label trial to assess the efficacy, safety, pharmacokinetics, and pharmacodynamics of dasiglucagon when administered as a rescue therapy for severe hypoglycemia in pediatric patients below 6 years of age with Type 1

Diabetes (T1D)

Protocol Version: Final 6.0, 12 Jul 2024

**Sponsor:** Zealand Pharma A/S

CVR No. DK 2004 5078 Sydmarken 11 DK-2860 Søborg

Denmark

Prepared by: Syneos Health

Albrechtstr.14, 80636 Munich, Germany

| Version | Date |
|---------|-----------------|
| V0.1 | 24 JUN 2022 |
| V0.2 | 08 JUL 2022 |
| V0.3 | 30 AUG 2022 |
| V1.0 | 31 AUG 2022 |
| V1.1 | 28 APR 2023 |
| V1.2 | 09AUG2023 |
| V1.3 | 18AUG2023 |
| V1.4 | 22AUG2023 |
| V.2.0 | 25AUG2023 |
| V.2.1 | 12SEP2024 |
| V.2.2 | 17DEC2024 |
| V.3.0 | 02JAN2025 Final |




## Approval

Upon review of this document, including the table, listing, and figure shells, the undersigned approves the statistical analysis plan. The analysis methods and data presentation are acceptable.

| Signature | Date |
|------------------------------|------|
| Syneos Health | |
| MSc, Principal Statistician, | |
| Zealand Pharma A/S | |
| MD, | |
| Zealand Pharma A/S | |
| Zealand Pharma A/S | |




# **Revision History**

| Version | Change |
|---|---|
| Version 2.0 | Statistical Analysis Plan updated to Protocol, version 4.0, 09 Mar 2023. |
| Version 3.0 | Statistical Analysis Plan updated to Protocol, version 6.0, 12 Jul 2024. Update of some shells based on dry-run comments. Addition of plots for plasma Glucose concentrations. Addition of a sensitivity analysis using the nominal predose time point as baseline. |




# TABLE OF CONTENTS

| 7 | ΓAΙ | BLE OF CONTENTS | 4 |
|---|---|---|---|
| LIS | ST ( | OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 7 |
| 1. | Π | NTRODUCTION | 8 |
| 2. | S | TUDY DOCUMENTS | 8 |
| 3. | S | TUDY OBJECTIVES | 8 |
| 4. | S | TUDY DESIGN AND PLAN | 8 |
| 5. | | DETERMINATION OF SAMPLE SIZE | |
| 6. | | GENERAL ANALYSIS CONSIDERATIONS | |
| 7. | | NOTATION OF TREATMENT GROUPS AND VISITS | |
| | | ANALYSIS SETS | |
| 8. | | | |
| 9. | | TUDY POPULATION | |
| | | Patient Disposition Protocol Deviations | |
| | 9.3 | | |
| | 9.4 | č , | |
| | | Medical History | 14 |
| 9 | 9.6 | Prior and Concomitant Medications and Current Diabetes Treatment | 14 |
| 10. | E | EFFICACY ANALYSES | 14 |
| ] | 10.1 | l Efficacy Variables | 15 |
| | | 2 Baseline Values | |
| 1 | 10.3 | 3 Adjustments for Covariates | 15 |
| | | 4 Handling of Dropouts or Missing Data | |
| | | 5 Interim Analysis and Data Monitoring | |
| | | 6 Examination of Subgroups | |
| | | 7 Multiple Comparison/Multiplicity | |
| | | 8 Multicenter Studies | |
| 11. | N | METHODS OF EFFICACY ANALYSIS | 16 |
| 1 | 11.1 | 1 Primary Efficacy Analyses | 16 |
| | | 2 Secondary Efficacy Analyses | |
| ] | 11.3 | 3 Further Efficacy Analyses | 16 |
| 12. | P | PHARMACOKINETIC ANALYSES | 16 |
| 1 | 12.1 | l Pharmacokinetic Variables | 16 |
| | | 2 Data Handling | |
| | | 3 Presentation of Plasma Concentrations | |

| | and Pharma<br>207-21052 | | Statistical Analysis Plan<br>2-Jan-25 |
|---|---|---|---|
| | | nination and Analysis of Pharmacokinetic Parameters | 20 |
| 13. | PHARM | ACODYNAMIC ENDPOINTS | 20 |
| 14. | SAFETY | ANALYSES | 21 |
| 1 | 4.1 Extent | of Exposure | 21 |
| | 14.1.1 | Diabetes Treatment prior hypoglycemia induction | |
| | 14.1.2 | Hypoglycemia Induction Procedure | |
| | 14.1.3 | Study Drug Administration | |
| 1 | 4.2 Local | Folerability | |
| | | se Events | |
| | 14.3.1 | Summary of Adverse Events | 23 |
| | 14.3.2 | Adverse Events by SOC and PT Terms | |
| 1 | 4.4 Clinica | ıl Laboratory Evaluation | |
| | | igns | |
| 1 | 4.6 Physic | al Examination | 24 |
| | - | ocardiogram | |
| | | nd Drink Intake | |
| | | uous Glucose Monitoring | |
| | | lucose Analyzer Data | |
| 1 | | nmunogenicity | |
| 15. | | ES TO PROTOCOL-SPECIFIED ANALYSES | |
| 16. | REFERE | NCES | 26 |
| | | ICES | |
| | | : PRESENTATION OF DATA AND PROGRAMMING SPE | |
| | _ | | |
| Ţ | astings | | 28 |
| | | Incomplete Dates (ie, Adverse Events and Concomitant Medicalculations | |
| | | ELIST OF TABLES, LISTINGS, AND FIGURES | |
| | | ction 14 | |
| | | ctions 16.1.2 | |
| AP | PENDIX C | : TABLE, FIGURE, LISTING LAYOUTS | 37 |
| Δ | nnendiy ( | 1: Study-Specific Shells for Section 14 | 38 |
| | | graphic Data | |
| | | ry Data | |
| | | ary Efficacy Endpoint | |
| | | ndary Efficacy Endpointndary Efficacy Endpoint | |
| | | oratory Analysis | |
| | | macokinetic Data | |
| | | Data | |
| 1 | T.J Salety | Data | |



| Zealand Pharma A/S | Statistical Analysis Plan |
|---|---|
| ZP4207-21052 | 2-Jan-25 |
| 14.3.1 Adverse Events | 69 |
| 14.3.2 Listings of Deaths, Other Serious and Significant Adverse Event | ts82 |
| 14.3.4 Abnormal Laboratory Value Listing (Each Patient) | 87 |
| 14.3.5 Extent of Exposure | 89 |
| 14.3.6 Other Safety Data | |
| Appendix C2: Study-Specific Shells for Section 16.2 | |
| 16.2. Patient Data Listings | |
| 16.2.1 Discontinued Patients | 107 |
| 16.2.2 Protocol Deviations | 109 |
| 16.2.3 Patients Excluded from the Analysis | 113 |
| 16.2.4 Demographic Data | |
| 16.2.5 Compliance and/or Drug Concentration Data | |
| 16.2.6 Individual Efficacy Response Data | 130 |
| 16.2.7 Adverse Event Listings | |
| 16.2.8 Listing of Individual Laboratory Measurements by Subject, Who | en Required by |
| Regulatory Authorities | 141 |
| 16.2.9 Other Data | |



## LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|---|---|
| ADA | anti-drug antibody |
| AE | adverse event |
| AESI | adverse event of special interest |
| ATC | anatomical therapeutic chemical |
| BMI | body mass index |
| CI | confidence interval |
| CSR | clinical study report |
| CGM | continuous glucose monitoring |
| CV | coefficient of variation |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| FAS | full analysis set |
| ICH | International Council for Harmonisation of Technical Requirements |
| | for Pharmaceuticals for Human Use |
| IMP | investigational medicinal product |
| IV | intravenous |
| BLOQ | below the limit of quantification |
| MDI | multiple daily injections |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PAS | PK analysis set |
| PD | pharmacodynamic(s) |
| PK | pharmacokinetic(s) |
| PT | preferred term |
| QTc | corrected QT interval |
| QTcF | corrected QT interval according to Fridericia's formula |
| SAE | serious adverse event |
| SAF | safety analysis set |
| SAP | statistical analysis plan |
| SC | subcutaneous |
| SD | standard deviation |
| SOC | system organ class |
| TEAE | treatment-emergent adverse event |
| TLFs | tables, listings, and figures |
| WHO | World Health Organization |




#### 1. INTRODUCTION

ZP4207-21052

This document outlines the statistical methods to be implemented during the analyses of data collected within the scope of Study ZP4207-21052, entitled "A Phase 3, single-administration open-label trial to assess the efficacy, safety, pharmacokinetics, and pharmacodynamics of dasiglucagon when administered as a rescue therapy for severe hypoglycemia in pediatric patients below 6 years of age with Type 1 Diabetes (T1D)". The purpose of this SAP is to provide specific guidelines for the statistical analyses. Any deviations from this plan will be documented in the CSR.

### 2. STUDY DOCUMENTS

The following study documents are used for the preparation of the SAP:

- Protocol, version 6.0, 12 Jul 2024
- Annotated electronic case report form (eCRF), version 6, 14Aug 2024
- Data management plan, version 3, 22 May 2024

### 3. STUDY OBJECTIVES

The primary study objective is:

- To assess the efficacy of dasiglucagon injection in children < 6 years of age with T1D</li>
   Other study objectives are as follows:
  - To assess PK of dasiglucagon in children with T1D
  - To assess the safety profile of dasiglucagon in children with T1D

#### 4. STUDY DESIGN AND PLAN

This trial will use a single-administration, open-label trial design to assess the ability of a single SC injection of dasiglucagon to increase plasma glucose in pediatric children with T1D with hypoglycemia. A total of 8 children will be included; 4 children receiving a dose of 0.3 mg and 4 children receiving a dose of 0.6 mg. Of the 4 children receiving 0.3 mg, at least 2 children must be below 2 years at screening. The remaining 2 children aged 2 years or above receiving 0.3 mg should preferably be below 4 years at screening. For children receiving the 0.6 mg dose, all must be above 2 years at screening. Before an eligible child is dosed, the dose level (0.6 mg or 0.3 mg) must be confirmed by the sponsor. Each child will be dosed after the safety assessment of the preceding child has been completed and assessed by the Trial Safety Group.

The trial will include the following visits (as illustrated in Figure 4-1).

- A screening visit (Visit 1, pre-treatment visit) in the period from Day -50 to Day -29
- A dosing visit (Visit 2), Day 1 (day of single dosing with IMP)
- A Safety follow-up visit (Visit 3) at Day 29 +5 days (the end-of-trial visit)

The primary endpoint of the trial is plasma glucose change from baseline at 30 minutes after IMP injection or at the time of rescue by IV glucose. Pharmacodynamics (PD) i.e., plasma glucose




will be assessed at baseline and 15 and 30 minutes after dosing, while the glucose levels will be monitored by CGM and by a plasma glucose analyzer during the dosing visit (Visit 2). PK will be assessed throughout a 300-minute period at the dosing visit (Visit 2). Safety will be assessed prior to dosing and throughout a 300-minute period after dosing and again at the follow-up visit. All data must be logged in the electronic case report form (eCRF).

Figure 4-1 Trial Design, taken from study protocol.





The schedule of assessments and trial procedures is available in the protocol.

The end of the trial is defined as the date of the last visit of the last patient in the trial. A patient is considered to have completed the trial if he/she has completed all phases of the trial including the last follow-up visit (Visit 3).

### 5. DETERMINATION OF SAMPLE SIZE

Eight children will be treated in this trial. The number of children is not based on a formal sample size calculation, evaluating the power of the trial, however some considerations have been made with respect to the precision of the estimate of the primary endpoint. In a previous pediatric trial with dasiglucagon (Trial ZP4207-17086), the mean plasma glucose change from baseline at 30 minutes after IMP injection was 96 mg/dL with a standard deviation (SD) of 20 mg/dL in children aged 6 to 11 years. Assuming the variation is the same in children < 6 years






Zealand Pharma A/S ZP4207-21052

of age, a 95% confidence interval will have a width of  $\pm$  25 mg/dL around the mean plasma glucose change with 95% probability, when 8 children are treated.

The power procedure in SAS with the onesamplemeans statement have been applied for the sample size consideration.

#### 6. GENERAL ANALYSIS CONSIDERATIONS

The statistical analyses will be reported using TLFs. The International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) numbering convention will be used for all TLFs.

Continuous variables will be summarized by presenting the number of observations, means, SDs, medians, minimums, and maximums. In addition, 95% confidence intervals (based on a *t* distribution if not otherwise stated) will be calculated if appropriate and detailed in the table shells. For logarithm-transformed data (relevant for selected PK summaries), the geometric mean and coefficient of variation % will also be provided.

Categorical variables will be summarized by presenting counts and percentages of subjects in corresponding categories. All possible categories as defined in the CRF should be populated, even if they have zero counts. Percentages for missing values are omitted and do not account for the percent calculation of other categories. Percentages are based on the total category count excluding the missing category if not otherwise mentioned. In certain tables (eg, AEs), the total number of subjects is used as the denominator. Footnotes will specify the percent basis in those cases.

All data collected in this trial and documented in the eCRFs will be presented in data listings. In case of termination of the trial, all data collected up to that time point will be included in the analysis.

All summary tables will be presented for the two treatment groups and total.

Individual subject data obtained from the eCRFs, external vendors, central clinical laboratory, central ECG laboratory, PK data, and any derived data will be presented by subject in data listings.

The analyses described in this plan are considered a priori, in that they have been defined before first patient dosed in the study. Any analyses performed after first patient dosed will be considered post hoc and exploratory. Post hoc analyses will be labeled as such on the output and identified in the CSR.

All analyses and tabulations will be performed using SAS® statistical software, version 9.4 or higher (SAS Institute Inc., Cary, North Carolina, USA). PK and PD analyses will be performed using Phoenix® WinNonlin®, version 8.3.4 or higher (Certara USA, Inc., Princeton, New Jersey, USA). This software was validated by Syneos Health in compliance with US 21 CFR Part 11 Regulation.




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 2-Jan-25

All statistical analysis will be performed as per Syneos SOPs.




### 7. NOTATION OF TREATMENT GROUPS AND VISITS

### **Notation of Treatment Groups**

The following notation of treatment groups will be used throughout the report:

| Full notation (as used in the study protocol) | Notation used throughout all tables, listings, and figures |
|---|---|
| dasiglucagon, 0.6 mg/0.6 mL SC injection | dasiglucagon 0.6mg |
| dasiglucagon, 0.3 mg/0.3mL SC injection | dasiglucagon 0.3mg |

Visit Terminology

| Visit | Notation used throughout all tables, listings, and figures |
|---|---|
| Screening VISIT 1 | Screening |
| Visit 2 (DOSING) | Dosing |
| Visit 3 (FOLLOW-UP) | Follow-up |

### **Study Days**

Study days corresponding to measurements are calculated as:

- Assessment date date of exposure to treatment + 1 (if assessment date is on or after the date of exposure to treatment).
- Assessment date date of exposure to treatment (if assessment date is before the date of
  exposure to treatment).

#### 8. ANALYSIS SETS

For the purposes of analysis, the following analysis sets are defined:

- Safety analysis set (SAF): All patients who were enrolled and received at least 1 dose of IMP.
- Full analysis set (FAS): All patients of the SAF.
- PK analysis set (PAS): All patients with at least one quantifiable plasma concentration.

Note: "Enrolled" requires parent's/legal guardian's agreement for the child to participate in a clinical trial following completion of the informed consent process and further that the child is screened and found eligible for the trial.

"Screened" requires a patient completed the informed consent process, regardless of whether the patient is eligible or not.

Data from these patients will be listed.




### 9. STUDY POPULATION

### 9.1 Patient Disposition

Patient disposition information will be summarized for all patients. Summaries will include the number of patients screened, enrolled, in each analysis set, completing/discontinuing the study and the primary reason for discontinuation.

#### 9.2 Protocol Deviations

Protocol deviations are collected according to the protocol deviation management plan. Major protocol deviations that could potentially affect the efficacy or safety conclusions of the study will be identified before database lock.

The final determination of major protocol deviations will be made during the data review meeting.

All protocol deviations, including the deviation designation (major or minor), and category will be presented in a data listing. Tables will be created for the SAF for all protocol deviations, summarized by the number of subjects in each deviation designation (major or minor) and category.

Due to the COVID-19 pandemic, the following additional analyses will be necessary. If a protocol deviation occurs, it will be documented if there is a relation to the COVID-19 pandemic. These COVID-19-related protocol deviations will be separately presented in tables as described above. In addition, the COVID-19-related protocol deviations will be listed.

### 9.3 Eligibility

A listing of subjects not fulfilling at least one eligibility criteria will be created.

### 9.4 Demographic and Baseline Characteristics

Demographic variables include age on consent date, sex, ethnicity, and race.

Other baseline characteristics include height, weight and BMI.

Descriptive statistics will be presented for age, age group (< 2 years, 2 to < 4 years, 4 to < 6 years), height, weight group (<15kg, >= 15kg) and BMI. Frequency counts and percentages will be presented for sex, ethnicity and race. Demographic and baseline characteristics will be summarized for the SAF.

Time since diagnosis of diabetes (date of informed consent – date of diabetes diagnosis + 1) in months will also be included in this summary, using descriptive statistics. If the day of diabetes diagnosis is not available, the calculation of duration will be based on month and year only, imputing the start day to 1. In case only the year is available, the start day will be imputed to be 1 and the start month will be imputed to be January.

A demographic and baseline characteristics listing will also be provided for the SAF.




### 9.5 Medical History

The verbatim term of the medical history condition/event will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 24.1.

A summary table will be prepared, summarizing the counts for each SOC and PT, ordered by descending order of incidence of SOC and PT.

A listing will be provided for the SAF.

#### 9.6 Prior and Concomitant Medications and Current Diabetes Treatment

Prior and concomitant medication and current diabetes treatment verbatim terms in the eCRFs will be mapped to the WHO Anatomical Therapeutic Chemical (ATC) classification and preferred names using the WHODrug dictionary, Global B3 format, Sep.1.2021 release.

The distinction between prior and concomitant medications is as follows:

- Prior medication are all medications which stopped before the first IMP administration during the study, regardless of start date.
- Concomitant medication is all medication that started prior to the first IMP administration
  and is still ongoing or stopped at the date of first study drug intake or medication that
  started on or after the date of the first IMP administration.
- If the start or stop date is incomplete and the allocation to prior or concomitant is unclear, the medication will be considered concomitant.

Partial dates will be imputed. For details on imputation rules, refer to Appendix A: Presentation of Data and Programming Specifications. Imputed dates are only used for classification of a medication as a prior or concomitant medication; no other calculation, such as durations, will be done.

Prior and concomitant medications and current diabetes treatment will be summarized by WHO ATC class (level 2) and preferred name. These summaries will present the number and percentage of patients using each medication. Patients may have more than 1 medication per ATC class and preferred name. At each level of patient summarization, a patient is counted once if they reported 1 or more medications at that level. Each summary will be ordered by descending order of incidence of ATC class and preferred name.

A listing will be created, listing all prior and concomitant medications as documented on the eCRF. A flag will be included in this listing, identifying which medications are prior and which are concomitant. An additional listing will be produced, listing all data collected on current diabetes treatment, as documented on the eCRF.

#### 10. EFFICACY ANALYSES

The primary efficacy analysis will be based on the FAS.




### 10.1 Efficacy Variables

The primary efficacy variable is:

 Plasma glucose concentration change from baseline at 30 minutes after IMP injection or at the time of rescue by IV glucose, if before 30 minutes.

The secondary efficacy variable is:

 Plasma glucose concentration change from baseline at 15 minutes after IMP injection or at the time of rescue by IV glucose, if before 15 minutes.

#### 10.2 Baseline Values

Unless otherwise noted, baseline is defined as the last non-missing value recorded prior to the first dose of study drug. Unscheduled visits will be used in the determination of baseline values, when applicable.

### 10.3 Adjustments for Covariates

No adjustments for covariates will be made.

### 10.4 Handling of Dropouts or Missing Data

No imputations will be made for missing values. Summaries will be based on observed data only. For handling of PK concentrations and results BLOQ, please refer to section 0

### 10.5 Interim Analysis and Data Monitoring

No interim analysis is planned for this study.

Data monitoring will be completed by the Trial Safety Group. New patients will only be dosed after safety assessment of the dosing visit for the preceding patient is completed and assessed by the Trial Safety Group. Thus, except for the first patient being dosed in the trial, investigators need written permission (eg, via an email) from the TSG chair to dose a patient in the trial.

More information on the TSG is available in the protocol.

### 10.6 Examination of Subgroups

No subgroup analysis is planned for this study.

#### 10.7 Multiple Comparison/Multiplicity

No adjustments for multiplicity will be made in this study.

#### 10.8 Multicenter Studies

This is a multicenter study with 8 subjects to be treated.


The expected low number of subjects per centers does not allow to do subgroup analysis within each site or to stratify by center.

#### 11. METHODS OF EFFICACY ANALYSIS

### 11.1 Primary Efficacy Analyses

The primary efficacy endpoint, plasma glucose change from baseline at 30 minutes after trial product injection or at the time of rescue by IV glucose if before 30 minutes, will be summarized using descriptive statistics and 95% confidence intervals (based on a *t* distribution).

### 11.2 Secondary Efficacy Analyses

The secondary efficacy endpoint, plasma glucose change from baseline at 15 minutes after IMP injection or at the time of rescue by IV glucose if before 15 minutes, will be summarized using descriptive statistics.

### 11.3 Further Efficacy Analyses

Untransformed and change from baseline plasma glucose at all timepoints, will be summarized using descriptive statistics.

A plot of mean glucose concentrations (untransformed) versus each time point will be provide and presented with error bars representing the Standard error of means (SEM).

A overlay plot of individual glucose concentrations (untransformed) versus each time point will be created.

A sensitivity analysis will be performed using the nominal pre-dose time point as baseline instead of the last valid measurement prior dosing.

#### 12. PPHARMACOKINETIC ANALYSES

The pharmacokinetic analysis will be based on the PAS set.

#### 12.1 Pharmacokinetic Variables

The following PK parameters for the dasiglucagon plasma concentrations will be estimated by non-compartmental analysis (NCA):

| PK parameter abbreviation | PK parameter | Calculation |
|---|---|---|
| AUC <sub>0-30min</sub> | Area under the plasma<br>concentration versus time curve<br>(AUC) from 0 to 30 minutes<br>post-dose | Linear trapezoidal rule for the ascending part of the concentration-time curve, logarithmic trapezoidal rule for the descending part. |




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 2-Jan-25

| PK parameter abbreviation | PK parameter | Calculation |
|---|---|---|
| AUC <sub>0-300min</sub> | AUC from 0 to 300 minutes post-dose | Linear trapezoidal rule for the ascending part of the concentration-time curve, logarithmic trapezoidal rule for the descending part. |
| AUC0-t | AUC from 0 to the last time point with a measured concentration Linear trapezoidal rule for the part of the concentration-time logarithmic trapezoidal rule for descending part. | |
| AUC <sub>0-inf</sub> | AUC from 0 to infinity post-dose | $(AUClast + Clast_{obs})/\lambda_{z,}$ where $Clast_{obs}$ is the concentration corresponding to Tlast (time of last measurable (positive) concentration). |
| C <sub>max</sub> | Maximum observed concentration | Taken directly from analytical data, selected from individual concentration data. The time when the first occurrence of Cmax is taken as Tmax. |
| $T_{\text{max}}$ | Time to C <sub>max</sub> | Taken directly from analytical data, selected from individual concentration data |
| λz | Terminal elimination rate constant of plasma dasiglucagon | Calculated by linear regression of the terminal linear portion of the log concentration vs. time curve. At least 3 concentrations in the terminal elimination phase will be required to calculate λz. |
| t <sub>1/2</sub> | Terminal plasma elimination half-life of dasiglucagon | $\operatorname{Ln}(2)/\lambda_{\mathbf{z}}$ |
| CL/f | Total body clearance of plasma dasiglucagon | Dose/ AUC <sub>0-inf</sub> |
| Vz/f | Volume of distribution of plasma dasiglucagon | Dose/ $(\lambda_z * AUC_{0-inf})$ or $CL/f/\lambda_z$ |
| MRT | Mean residence time of plasma<br>dasiglucagon | AUMCinf/ AUC <sub>0-inf</sub> where AUMCinf is the area under the first moment curve as estimated by WinNonlin. |




## 12.2 Data Handling

Refer to **Table 12-1** for details on which PD and PK samples to be collected based on body weight at Visit 1 and Visit 2.

Table 12-1 PD (for efficacy) and PK Sampling Based on Body Weight

| Body weight at Visit 2 | Visit 2 | |
|--------------------------------|--------------------|--------------------|
| | PD samples to draw | PK samples to draw |
| BW> 10.0 kg | pre-dose | pre-dose |
| | 15 min | 10 min |
| | 30 min | 20 min |
| | | 30 min |
| | | 40 min |
| | | 60 min |
| | | 90 min |
| | | 140 min |
| | | 220 min |
| | | 300 min |
| $10.0 \ge BW > 9.0 \text{ kg}$ | pre-dose | pre-dose |
| | 15 min | 10 min |
| | 30 min | 20 min |
| | | 30 min |
| | | 40 min |
| | | 60 min |
| | | 90 min |
| | | 140 min |
| | | 300 min |
| $9.0 \ge BW > 8.0 \text{ kg}$ | pre-dose | pre-dose |
| | 30 min | 10 min |
| | | 20 min |
| | | 30 min |
| | | 40 min |
| | | 60 min |
| | | 90 min |
| | | 140 min |
| | | 300 min |

Abbreviations: BW=body weight; PD=pharmacodynamics; PK=pharmacokinetics

The raw plasma concentration data will be handled as follows:

### For summary tables and figures for plasma concentrations:

- i.) For all pre-dose samples, the sampling time will be set to zero.
- ii.) For post-dose samples, the planned sampling time will be used in summary tables, and the actual sampling times will be used for all figures of individual concentrations.
- iii.) All concentration values below the Limit of Quantification (BLOQ) will be set to zero.
- iv.) Missing post-dose values will not be replaced.


### For determination of PK metrics:

- *i.)* For all pre-dose samples, the sampling time will be set to zero.
- ii.) For post-dose samples, the actual sampling time will be used.
- iii.) All pre-dose concentration values will be set to zero.
- iv.) Post-dose concentration values BLOQ after  $T_{max}$  will be set to missing.
- v.) Missing post-dose values will not be replaced.
- vi.) A concentration that is BLOQ is assigned a value of zero if it occurs in a profile after dosing at time zero and before the first measurable concentration.
- vii.) If a BLOQ value occurs after a measurable concentration in a profile and is followed by a value above the lower limit of quantification, then the BLOQ is treated as missing data, and the time point is ignored in the computations.
- viii.) If a BLOQ value occurs at the end of the collection interval (after the last quantifiable concentration) it is treated as missing data.
- ix.) If two BLOQ values occur in succession after Cmax, the profile is deemed to have terminated at the first BLOQ value and any subsequent concentrations and time points are omitted from pharmacokinetic calculations.

### 12.3 Presentation of Plasma Concentrations

### Individual plasma concentration results:

A raw data listing will be provided displaying the dasiglucagon concentration as reported and nominal and actual sampling times relative to the start dose of study drug. Results will be displayed using 3 significant digits.

### Summary statistics of plasma concentrations:

The dasiglucagon plasma concentrations will be summarized using descriptive statistics (n, arithmetic mean, SD, coefficient of variation (CV) % of arithmetic mean, median, minimum, maximum, geometric mean, and CV % for the geometric mean).

Results will be displayed using 3 significant digits.

The CV % for the geometric mean will be calculated using the following formula:

$$CV$$
 (%) =  $100 * \sqrt{e^{SD^2} - 1}$ 

Where SD is of the natural-log transformed data.

### Figures:

Individual and mean concentration-time profiles will be provided on linear and semilogarithmic scales. For individual concentration-time profiles, the actual sampling times will be used.




Zealand Pharma A/S Statistical Analysis Plan
ZP4207-21052 2-Jan-25

Mean concentration-time profiles will be provided on linear and semilogarithmic scales and may be presented with error bars representing the Standard error of means (SEM).

### 12.4 Determination and Analysis of Pharmacokinetic Parameters

Full precision concentration data and actual sample times will be used for the determination of all PK parameters.

Raw plasma concentrations for the derivation of PK parameters will be handled as described in Section 12.1.

The PK parameters as listed in Section 12.1 will be estimated.

### Reporting of missing PK parameters:

The percentage of extrapolated AUC should not exceed 20% of AUC<sub>inf</sub> for each individual profile. If the percentage of extrapolated AUC is more than 20%, the individual AUC<sub>inf</sub> result and parameters depending on AUC<sub>inf</sub> will be listed but flagged as not reliably calculated. They will generally not be included in descriptive statistics and statistical testing procedures.

The terminal half-life regression analysis should contain data from at least 3 different time points after  $C_{max}$  in the terminal phase and as many data points as possible (always including the last quantifiable concentration but excluding the concentration at  $T_{max}$ ), consistent with the assessment of a straight line on the log-transformed scale. The coefficient of regression ( $r^2$ ) should be larger than or equal to 0.80. If at least one of these conditions is not fulfilled, the terminal half-life and parameters depending on  $t_{1/2}$  will be listed but flagged as not reliably calculated. They will generally be excluded from descriptive statistics and statistical testing procedures. However, if the reliability of the estimated terminal half-life is judged to be reasonable by the pharmacokineticist who oversees the PK analysis, the  $t_{1/2}$  and related parameters would not be excluded.

### Individual PK parameters:

A raw data listing will be provided displaying the individual PK parameters. Results will be displayed using 3 significant digits.

### **Summary statistics of PK parameters:**

Pharmacokinetic parameters will be summarized using descriptive statistics (n, arithmetic mean, SD, CV% for the arithmetic mean, median, minimum, maximum, geometric mean, and CV% for the geometric mean). The geometric mean and CV% for the geometric mean will not be calculated for  $T_{\text{max}}$ . Results will be displayed using 3 significant digits.

#### 13. PHARMACODYNAMIC ENDPOINTS

Pharmacodynamic endpoints coincide with the primary and secondary efficacy endpoints. The plasma glucose profile for assessment of the primary and secondary clinical efficacy endpoints will be assessed based on plasma glucose concentration data from samples collected at the dosing visit (Visit 2).




Plasma glucose is determined at pre-dose and at 15 and 30 minutes after dosing. The actual time of blood sampling should not deviate from the nominal time by more than  $\pm$  1 minute for the collection time points. Pre-dose is defined as within 2 minutes prior to dosing.

#### 14. SAFETY ANALYSES

All safety analyses will be based on the SAF.

### 14.1 Extent of Exposure

### 14.1.1 Diabetes Treatment prior hypoglycemia induction

A summary table will be prepared showing the number (percentage) of patients who used any of the following:

- MDI
- Insulin pump

All details related to the diabetes treatment prior hypoglycemia induction will be provided in a listing.

### 14.1.2 Hypoglycemia Induction Procedure

A summary table will be prepared summarizing the data collected for the hypoglycemia induction procedure. Frequency counts and percentages will be presented for the number of patients where the hypoglycemia induction procedure was performed and for the number of patients where glucose was administered intravenously prior to dosing.

The duration in minutes between stop of insulin pump (respectively for multiple daily injections (MDI) users, last basal dose before the Hypoglycaemia procedure) and time when Hypoglycaemia procedure was initiated will be calculated and summarized.

Descriptive statistics will be given for the total amount of insulin administered to induce hypoglycemia and the total amount of glucose administered during the induction procedure.

All details related to the hypoglycemia induction procedure will be provided in a listing.

### 14.1.3 Study Drug Administration

All data related to study drug administration will be provided in a data listing.

### 14.2 Local Tolerability

Local tolerability assessments at 30, 120, and 300 minutes after IMP administration will be performed to assess the following:




#### Zealand Pharma A/S ZP4207-21052

- Spontaneous pain
- Pain on palpation
- Itching
- Redness
- Edema
- Induration/infiltration
- Other reaction

Injection site reactions and any findings will be reported as AEs.

The analysis of local tolerability will include a summary table displaying the counts and percentages of patients experiencing local symptoms by time point, symptom and severity. Additionally, all details collected from the local tolerability assessments will be provided in a data listing. Any "other types of reaction" will be summarized under the umbrella term "Other".

#### 14.3 Adverse Events

Unless otherwise stated, all AE summary tables will be restricted to TEAEs, which are defined as those AEs that occurred after dosing and those existing AEs that worsened during the study. Partial dates will be imputed. For details on imputation rules, refer to Appendix A: Presentation of Data and Programming Specifications. Imputed dates are only used to determine if an AE is a TEAE: no other calculation, such as durations, will be done. If it cannot be determined whether the AE is treatment-emergent due to a partial onset date, then it will be counted as treatment-emergent. Verbatim terms in the eCRFs will be mapped to SOCs and PTs using MedDRA, version 24.1.

TEAE summaries that are displayed by SOC and PT, will be ordered by descending patient count, by SOC and PT.

### Causal relationships

Causal relationship between the occurrence of an AE and the administration of the study drug is assessed by the investigator according to classification scheme: 0=not related, 1=unlikely, 2=possible and 3=probable. Probable and possible relationships will be included under the category related. All AEs must have a causal relationship assigned. In case of a missing relationship, a query will be raised in order to obtain causality assessment. In case no clarification of relationship via query is possible the missing relationship will be set to related for the analysis.

### Severity

Severity grading will differ between 1=mild, 2=moderate and 3=severe. For AEs having a missing severity, the severity will not be imputed and kept as missing.




### 14.3.1 Summary of Adverse Events

A summary table of all AEs will be prepared, summarizing the number and percentage of patients with at least 1 AE and the total number of AEs in the following categories:

- AEs that occurred during screening
- 2. TEAEs
- 3. TEAEs occurring within 12 hours after dosing
- 4. TEAEs, which are AESIs
- 5. TEAEs, which are an other important event
- 6. TEAEs, which are injection site reactions based on investigator assessment on the eCRF
- IMP related TEAEs
- 8. TEAEs, which are SAEs
- IMP related TEAEs, which are SAEs
- 10. Deaths

### 14.3.2 Adverse Events by SOC and PT Terms

The analysis of AEs will include summary tables displaying the counts and percentages of patients experiencing AEs by SOC and PT. If a patient has more than 1 AE which codes to the same PT, the patient will be counted only once for that PT. The total number of events documented per SOC and PT will also be displayed. Summaries will be ordered by descending order of incidence of SOC and PT, within each SOC based on the frequency (proportion of patients) in the dasiglucagon group.

Frequency tables will be prepared by MedDRA terms (SOC and PT) summarizing the categories 1 to 9 as listed in Section 14.3.1.

All details relating to adverse events will also be provided in a data listing. Additional listings will be produced to display: AEs for screening failures, any AESIs, AEs leading to discontinuation of IMP, SAEs and any AEs leading to death.

### 14.4 Clinical Laboratory Evaluation

Laboratory parameters (clinical chemistry, hematology, coagulation) for continuous results will be summarized using descriptive statistics at baseline and at each post-baseline time point. Changes from baseline will also be summarized.

The numbers in each category (above/below/within the relevant reference ranges) will be counted and percentages presented for each laboratory test result at each scheduled visit.

Three separate listings will be produced, which will include all data related to clinical chemistry, hematology, and coagulation laboratory tests.




### 14.5 Vital Signs

Vital signs will be summarized using descriptive statistics at baseline and at each scheduled postbaseline visit and time point. Changes from baseline will also be summarized.

Categorical results for interpretation (normal/abnormal) will be summarized using frequency counts at baseline and at each scheduled post-baseline visit and time point.

All data related to vital signs will also be included in a data listing.

### 14.6 Physical Examination

Physical examination results will be included in data listings only.

### 14.7 Electrocardiogram

The following 12-lead ECG parameters will be summarized using descriptive statistics at screening.

- Heart Rate (beats/min)
- PR Interval (msec)
- QRS Interval (msec)
- QT Interval (msec)
- QTc Interval (msec)
- QTcF Interval (msec) [QTc calculated using Fredericia's formula]

Additionally, the number of patients with an ECG interpretation of normal/abnormal clinically significant/abnormal not clinically significant will be summarized at screening.

All ECG data will also be provided in a data listing.

#### 14.8 Food and Drink Intake

Data collected on the food and drink intake of patients at Visit 2 (pre-dose and post-dose) will be provided in a data listing only.

### 14.9 Continuous Glucose Monitoring

CGM data will be presented graphically as individual plots (per patient) of glucose measurements over time, from the time of stopping the participant's insulin pump to 300 minutes after dasiglucagon administration.

A secondary y-axis will be displayed to show Glucose measurements in mmol/L additionally to mg/dl. Results are converted into the unit 'mmol/L' by using the conversion factor 0.0555 (i.e. Glucose [mmol/L]=Glucose [mg/dl] \*0.0555).

All CGM data will also be included in a data listing.




### 14.10 Glucose Analyzer Data

Glucose Analyzer data will be summarized by time point and included in a data listing.

In addition, individual time-concentration curves will be created using the time of first dosing of IMP as relative starting point.

### 14.11 Immunogenicity

Occurrence of ADA will be analyzed descriptively. ADA and results from associated characterization assays will be presented descriptively.

ADA will be derived from the number of patients having an ADA-positive sample during the trial. Positive anti-dasiglucagon antibody samples from treatment-induced or treatment-boosted (titer increase above 4-fold) is defined as ADA-positive.

### 15. CHANGES TO PROTOCOL-SPECIFIED ANALYSES

No changes were made to the protocol-specified analysis.




Zealand Pharma A/S ZP4207-21052 Statistical Analysis Plan 2-Jan-25

### 16. REFERENCES

International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH). ICH Harmonised Tripartite Guideline. The clinical evaluation of QT/QTc interval prolongation and proarrhythmic potential for non-antiarrhythmic drugs E14. November 2005.




#### 17. APPENDICES

#### APPENDIX A: PRESENTATION OF DATA AND PROGRAMMING SPECIFICATIONS

#### General

- Specialized text styles, such as bold, italics, borders, shading, and superscripted and subscripted text will not be used in tables, figures, and data listings (TFLs) unless they add significant value to the TFL.
- Only standard keyboard characters are to be used in tables and data listings.
- Special characters, such as nonprintable control characters and printer- or font-specific characters, will not be used in a TFL.
- Hexadecimal character representations are allowed (eg, μ, α, and β).
- All footnotes will be left justified and at the bottom of a page. Footnotes must be used sparingly and add value to the TFL.

#### Tables

- Means and medians will be presented to 1 decimal place more than the raw data.
   Standard deviations will be presented to 2 decimal places more than the raw data.
   Minimums and maximums will be reported with the same number of decimal places as the raw data.
- Percentages will be presented to the tenths place.
- For frequency counts of categorical variables, categories whose counts are zero will be displayed for the sake of completeness. For example, if none of the subjects discontinue due to "lost to follow-up," this reason will be included in the table with a count of 0.
   Categories with zero counts will not have zero percentages displayed.
- Lower and upper CI values must be presented to 1 decimal place more than the raw/derived data (ie, to the same number of decimal places as the mean).
- Percentiles (eg, 25% and 75%) must be presented to 1 decimal place more than the raw/derived data.
- For all inferential analyses, P values will be rounded to 4 decimal places (or at the highest level of precision) with a leading zero (0.0001). P values less than 0.0001 will be presented as "<0.0001."</li>
- The last footnotes will be:
  - "Source: xxx", where xxx indicates the source table number(s), if applicable (in case aggregated results, such as the mean or median, are plotted), source listing(s) (in case individual responses are plotted), and/or source dataset(s) (eg, ADaM).
  - "PROGRAM SOURCE:...\xx.sas, DATA CUT-OFF DATE: DD Mmm YYYY, RUN DATE: DD Mmm YYYY hh:mm".




### **Figures**

- Legends will be used for all figures with more than 1 variable or item displayed.
- Figures will be in black and white but can be in color to add value to the clarity and readability of a figure. Lines must be wide enough to see the line after being copied.
- The last footnotes will be:
  - "Source: xxx", where xxx indicates the source listing number(s) and/or source dataset(s) (eg, ADaM).
  - "PROGRAM SOURCE:...\xx.sas, DATA CUT-OFF DATE: DD Mmm YYYY, RUN DATE: DD Mmm YYYY hh:mm".

### Listings

- If not otherwise specified, all data listings will be sorted by center, subject number, visit, and date/time, as appropriate.
- All date values will be presented in a SAS® statistical software, version 9.4 or higher (SAS Institute Inc) date format (eg, 29AUG2001).
- All observed time values will be presented using a 24-hour clock format (HH:MM:SS) (eg, 01:35:45 or 11:26). Seconds will only be reported if they were measured as part of the study.
- The last footnote will be "PROGRAM SOURCE:...\xx.sas, DATA CUT-OFF DATE: DD Mmm YYYY, RUN DATE: DD Mmm YYYY hh:mm".

### Missing or Incomplete Dates (ie, Adverse Events and Concomitant Medications)

The most conservative approach will be systematically considered. If the adverse event (AE) onset date is missing/incomplete, it is assumed to have occurred during the study treatment phase (ie, considered a treatment-emergent AE) except if the partial onset date or other data, such as the stop date, indicates differently. Similarly, a medication with partial start and stop dates could be considered as both a prior and concomitant medication.

The following algorithms will be applied to missing and incomplete start and stop dates:

### Start Dates

- If the day portion of the start date is missing, then the start date will be estimated to be
  equal to the date of the first dose of study drug, provided the start month and year are the
  same as the date of the first dose of study drug and stop date is either after the date of the
  first dose of study drug or completely missing. Otherwise, the missing day portion will be
  estimated as "01."
- If both the day and month portions of the start date are missing, then the start date will be
  estimated to be equal to the date of the first dose of study drug, provided the start year is
  the same as the date of the first dose of study drug and stop date is either after the date of






the first dose of study drug or completely missing. Otherwise, the event will be assumed to start on the first day of the given year (eg.,??-???-2013 is estimated as 01-JAN-2013).

• If the start date is completely missing and stop date is either after the date of the first dose of study drug or completely missing, then the start date will be estimated to be equal to the date of the first dose of study drug. Otherwise, the start date will be estimated to be the first day of the same year as the stop date. All other non-AE and non-concomitant medication day calculations where only partial dates are available will be handled as follows: the first day of the month will be used in the calculations if the day part of a start date is missing, and January 1 will be used if both the month and day parts of a start date are missing.

### Stop Dates

Zealand Pharma A/S

ZP4207-21052

- If only the day of resolution is unknown, the day of resolution of the event will be assumed to be the last day of the month (eg,??-JAN-2013 will be treated as 31-JAN-2013).
- If both the day and month of resolution are unknown, the day of resolution of the event will be assumed to be the last day of the year (eg,??-???-2013 will be treated as 31-DEC-2013).
- If the stop date of the event is completely missing or event is continuing, the event
  resolution will be assumed to be after the first dose of study drug, and the stop date will
  be imputed using the last known date on the study.

### **Standard Calculations**

Variables requiring calculation will be derived using the following formulas:

- Days: A duration expressed in days between 1 date (date1) and another later date (date2) is calculated using the following formula: duration in days = date2 date1 + 1
- Months: A duration expressed in months is calculated using the INTCK function of SAS using the following formula: months = intck('month', 'date1'd, date2'd, 'continuous')
- Years: A duration expressed in years between 1 date (date1) and another later date (date2) is calculated using the following formula: duration in years = intck('year', 'date1'd, 'date2'd, 'continuous')
- Body Mass Index (BMI): BMI is calculated using height and weight using and is calculated using the following formula: BMI (kg/m²) = weight (kg) / [[height (cm) / 100]²]
- Change from baseline: Change from baseline will be calculated using the following formula: change = analysis value (including the baseline value) baseline value




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 2-Jan-25

 Percent change from baseline: Percent change from baseline will be calculated using the following formula: percent change from baseline = (analysis value (including the baseline value) – baseline value)/baseline value × 1


Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

## APPENDIX B: LIST OF TABLES, LISTINGS, AND FIGURES

The following proposal for Sections 14 and 16.2 is completed according to ICH E3 guidelines The heading numbers and description are in **bold**. Minor changes from this planned index do not need to be amended in the SAP.

### **Index of Section 14**

| Table/Figure number | Table/Figure title | Analysis Set | Comment |
|---|---|---|---|
| 14 | Tables and Figures Referred to but not Included in the Text | | |
| 14.1 | Demographic Data | | |
| 14.1.1 | Patient Disposition | All Patients | |
| 14.1.2 | Patient Number by Country and Center | Safety Analysis Set | |
| 14.1.3 | Protocol Deviations | Safety Analysis Set | |
| 14.1.4 | COVID-19 Related Protocol Deviations | Safety Analysis Set | |
| 14.1.5 | Demographic and Baseline Characteristics | Safety Analysis Set | |
| 14.1.6 | Medical History | Safety Analysis Set | |
| 14.1.7 | Prior Medications | Safety Analysis Set | |
| 14.1.8 | Concomitant Medications | Safety Analysis Set | |
| 14.1.9 | Current Diabetes Treatment | Safety Analysis Set | |
| 14.2 | Efficacy Data | | |
| 14.2.1 | Primary Efficacy Endpoint | | |
| 14.2.1.1 | Plasma Glucose Change from Baseline at 30 minutes after IMP Injection | Full Analysis Set | |
| 14.2.2 | Secondary Efficacy Endpoint | | |
| 14.2.2.1 | Plasma Glucose Change from Baseline at 15 minutes after IMP Injection | Full Analysis Set | |
| 14.2.3 | Exploratory Analysis | | |
| 14.2.3.1 | Plasma Glucose Change from Baseline at 30 minutes after IMP Injection in Subjects Without Rescue IV Glucose | Full Analysis Set | |
| 14.2.3.2 | Plasma Glucose Change from Baseline at 15 minutes after IMP Injection in Subjects Without Rescue IV Glucose | Full Analysis Set | |
| 14.2.3.3 | Plasma Glucose - untransformed and change from baseline at each time point | Full Analysis Set | |




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
2-Jan-25

| P4207-21052 | | | 2-Jan- |
|---|---|---|---|
| 14.2.3.4 | Mean glucose concentrations versus time - original scale | Full Analysis Set | Figure |
| 14.2.3.5 | Individual glucose concentrations versus time - original scale | Full Analysis Set | Figure |
| 14.2.3.6 | Plasma Glucose Change from Baseline at 30 minutes after IMP Injection –<br>Sensitivity Analysis | Full Analysis Set | |
| 14.2.3.7 | Plasma Glucose Change from Baseline at 15 minutes after IMP Injection –<br>Sensitivity Analysis | Full Analysis Set | |
| 14.2.3.8 | Plasma Glucose - untransformed and change from baseline at each time point- Sensitivity Analysis | Full Analysis Set | |
| 14.2.4 | Pharmacokinetic Data | | |
| 14.2.4.1 | Descriptive Statistics for dasiglucagon Plasma Concentration | PK Analysis Set | |
| 14.2.4.2 | Mean dasiglucagon Concentration-time Profile – linear scale | PK Analysis Set | Figure |
| 14.2.4.3 | Mean dasiglucagon Concentration-time Profile – semi-log scale | PK Analysis Set | Figure |
| 14.2.4.4 | Individual dasiglucagon Concentration-time Profiles – linear scale | PK Analysis Set | Figure |
| 14.2.4.5 | Individual dasiglucagon Concentration-time Profiles – Semi-log scale | PK Analysis Set | Figure |
| 14.2.4.6 | Descriptive Statistics for PK Parameters | PK Analysis Set | |
| 4.3 | Safety Data | | |
| 14.3.1 | Adverse Events | | |
| 14.3.1.1 | Overall Summary of Adverse Events | Safety Analysis Set | |
| 14.3.1.2 | Treatment-Emergent Adverse Events by System Organ Class and Preferred Term | Safety Analysis Set | |
| 14.3.1.3 | Treatment-Emergent Adverse Events occurring within 12 hours after dosing by System Organ Class and Preferred Term | Safety Analysis Set | |
| 14.3.1.4 | Adverse Events that occurred during Screening, by System Organ Class and Preferred Term | Safety Analysis Set | |
| 14.3.1.5 | Treatment-Emergent Adverse Events of Special Interest, by System Organ Class and Preferred Term | Safety Analysis Set | |
| 14.3.1.6 | Treatment-Emergent Adverse Events that are Other Important Events, by<br>System Organ Class and Preferred Term | Safety Analysis Set | |
| 14.3.1.7 | Treatment-Emergent Adverse Events that are Injection Site Reactions, by<br>System Organ Class and Preferred Term | Safety Analysis Set | |
| 14.3.1.8 | Treatment-Emergent Adverse Events that are IMP Related, by System Organ Class and Preferred Term | Safety Analysis Set | |




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
2-Jan-25

| CP4207-21052 | | | 2-Jan-25 |
|---|---|---|---|
| 14.3.1.9 | Serious Treatment-Emergent Adverse Events, by System Organ Class<br>and Preferred Term | Safety Analysis Set | |
| 14.3.1.10 | Serious Treatment-Emergent Adverse Events that are IMP Related, by<br>System Organ Class and Preferred Term | Safety Analysis Set | |
| 14.3.1.11 | Local Tolerability Assessment | Safety Analysis Set | |
| 14.3.2 | Listings of Deaths, Other Serious and Significant Adverse Events | | |
| 14.3.2.1 | Serious Adverse Events | Safety Analysis Set | |
| 14.3.2.2 | Adverse Events Leading to Premature Discontinuation of Study Drug | Safety Analysis Set | |
| 14.3.2.3 | Adverse Events Leading to Death | Safety Analysis Set | |
| 14.3.3 | Narratives of Deaths, Other Serious and Certain Other Significant<br>Adverse Events | | This is a cross-reference to section 12.3.2 of the CSR |
| 14.3.4 | Abnormal Laboratory Value Listing (Each Patient) | | |
| 14.3.4.1 | Abnormal Laboratory Values | Safety Analysis Set | |
| 14.3.5 | Extent of Exposure | | |
| 14.3.5.1 | Diabetes Treatment Prior Hypoglycemia | Safety Analysis Set | |
| 14.3.5.2 | Hypoglycemia Induction Procedure | Safety Analysis Set | |
| 14.3.6 | Other Safety Data | | |
| 14.3.6.1 | Continuous Glucose Monitoring - Individual Glucose Concentration-time<br>Profiles | PK Analysis Set | Figure |
| 14.3.6.2 | Glucose Analyzer Data | Safety Analysis Set | |
| 14.3.6.2 | Laboratory Data | | |
| 14.3.6.2.1 | Hematology Results | Safety Analysis Set | |
| 14.3.6.2.2 | Hematology Results – Reference Range Analysis | Safety Analysis Set | |
| 14.3.6.2.3 | Chemistry Results | Safety Analysis Set | |
| 14.3.6.2.4 | Chemistry Results – Reference Range Analysis | Safety Analysis Set | |
| 14.3.6.2.5 | Coagulation Results | Safety Analysis Set | |
| 14.3.6.2.6 | Coagulation Results – Reference Range Analysis | Safety Analysis Set | |




Zealand Pharma A/S
Statistical Analysis Plan
ZP4207-21052
2-Jan-25

| 21 1207 21002 | | | 2 can 25 |
|---------------|----------------|---------------------|----------|
| 14.3.6.2.7 | Immunogenicity | Safety Analysis Set | |
| 14.3.6.3 | Vital Signs | Safety Analysis Set | |
| 14.3.6.4. | ECG Data | Safety Analysis Set | |

Abbreviations: ECG=electrocardiogram; ICH=International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use.




Zealand Pharma A/S ZP4207-21052

## **Index of Sections 16.1.2**

| ICH listing number | Listing title | Analysis Set | Comments |
|---|---|---|---|
| 16.2 | Patient Data Listings | | |
| 16.2.1 | Discontinued Patients | | |
| 16.2.1.1 | Patient Disposition | All Patients | |
| 16.2.2 | Protocol Deviations | | |
| 16.2.2.1 | Protocol Deviations | Safety Analysis Set | |
| 16.2.2.2 | COVID-19 Related Protocol Deviations | Safety Analysis Set | |
| 16.2.2.3 | Patients not Fulfilling at least one Inclusion/Exclusion Criteria | All Screened Patients | |
| 16.2.3 | Patients Excluded from the Analysis | | |
| 16.2.3.1 | Patients Excluded from Analysis | All Enrolled Patients | |
| 16.2.4 | Demographic Data | | |
| 16.2.4.1 | Demographic and Baseline Characteristics | Safety Analysis Set | |
| 16.2.4.2 | Medical History | Safety Analysis Set | |
| 16.2.4.3 | Prior and Concomitant Medications | Safety Analysis Set | |
| 16.2.4.4 | Current Diabetes Treatment | Safety Analysis Set | |
| 16.2.5 | Compliance and/or Drug Concentration Data | | |
| 16.2.5.1 | Study Drug Administration | Safety Analysis Set | |
| 16.2.5.2 | Diabetes treatment prior hypoglycemia induction - MDI user | Safety Analysis Set | |
| 16.2.5.3 | Diabetes treatment prior hypoglycemia induction - meal-time/ bolus insulins | Safety Analysis Set | |
| 16.2.5.4 | Diabetes treatment prior hypoglycemia induction - pump user | Safety Analysis Set | |
| 16.2.5.5 | Hypoglycemia Induction Procedure | Safety Analysis Set | |
| 16.2.5.6 | dasiglucagon Plasma Concentrations | Safety Analysis Set | |
| 16.2.5.7 | dasiglucagon PK Parameters | Safety Analysis Set | |
| 16.2.5.8 | Continuous Glucose Monitoring | Safety Analysis Set | |
| 16.2.6 | Individual Efficacy Response Data | | |
| 16.2.6.1 | Plasma Glucose Concentrations | Safety Analysis Set | |




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
2-Jan-25

| ZP4207-21052 | | 2-Jan-25 |
|---|---|---|
| 16.2.7 | Adverse Events Listings | |
| 16.2.7.1 | Adverse Events | Safety Analysis Set |
| 16.2.7.2 | Adverse Events of Special Interest | Safety Analysis Set |
| 16.2.7.3 | Hemodynamic Changes During Adverse Events of Special Interest | Safety Analysis Set |
| 16.2.7.4 | Other Important Events | Safety Analysis Set |
| 16.2.7.5 | Details of Other Important Events | Safety Analysis Set |
| 16.2.7.6 | Local Tolerability Assessment | Safety Analysis Set |
| 16.2.7.7 | Death details | Safety Analysis Set |
| 16.2.7.8 | Adverse Events for Screening Failures | Screening Failures |
| 16.2.8 | Listing of Individual Laboratory Measurements by Subject, When Required by Regulatory Authorities | |
| 16.2.8.1 | Hematology | Safety Analysis Set |
| 16.2.8.2 | Chemistry | Safety Analysis Set |
| 16.2.8.3 | Coagulation | Safety Analysis Set |
| 16.2.9 | Other Data | |
| 16.2.9.1 | Vital Signs | Safety Analysis Set |
| 16.2.9.2 | Physical Examination | Safety Analysis Set |
| 16.2.9.3 | Electrocardiogram | Safety Analysis Set |
| 16.2.9.4 | Hospitalization | Safety Analysis Set |
| 16.2.9.5 | Immunogenicity | Safety Analysis Set |
| 16.2.9.6 | Food and Drink Intake | Safety Analysis Set |
| 16.2.9.7 | Technical Complaints | Safety Analysis Set |

Abbreviations: ICH=International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use.



# APPENDIX C: TABLE, FIGURE, LISTING LAYOUTS

Table, Figure and Listing layouts (shells) are provided in a separate document.




Appendix C1: Study-Specific Shells for Section 14

14.1 Demographic Data




 Zealand Pharma A/S
 Statistical Analysis Plan

 ZP4207-21052
 2-Jan-25

 Zealand Pharma A/S
 Clinical Study Report

Protocol Number: ZP4207-21052

# Table 14.1.1 Patient Disposition All Patients

Page x of y

| | dasiglucagon 0.3mg | dasiglucagon 0.6mg | Total |
|---|---|---|---|
| Number of patients screened | | | xx |
| Number of patients enrolled[a] | xx | xx | xx |
| Number of patients in the Safety Analysis Set[b] | xx ( 100.0%) | xx ( 100.0%) | xx (100.0%) |
| Number of patients in the Full Analysis Set[c] | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Number of patients in the PK Analysis Set[d] | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Completed Study (based on Safety Analysis Set) | | | |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Primary reason for study discontinuation | | | |
| Adverse Event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Death | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Disease Relapse | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Failure to Meet Randomization criteria | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lack of Efficacy | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Lost to Follow-up | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Non-Compliance with Study Drug | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Physician Decision | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Progressive Disease | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Protocol Deviation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Recovery | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Screen Failure | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Site Terminated by Sponsor | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Study Terminated by Sponsor | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Technical Problems | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Withdrawal by Parent/Guardian | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Percentages are based on the total number of patients enrolled.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY hh:mm


<sup>[</sup>a] Requires parent's/legal guardian's agreement for the child to participate in a clinical trial following completion of the informed consent process and further that the child is screened and found eligible for the trial.

<sup>[</sup>b] All patients who were enrolled and received at least 1 dose of study drug.

<sup>[</sup>c] All patients of the safety analysis set.

<sup>[</sup>d] All patients with at least one quantifiable plasma concentration.



Programming Notes:

1) Include all discontinuation reasons (even if no subjects discontinued for that reason). Sort in order as on CRF.




Clinical Study Report Zealand Pharma A/S Protocol Number: ZP4207-21052

Page x of y

# Table 14.1.2 Patient Number by Country and Center Safety Analysis Set

| Center<br>Number | dasiglucagon 0.3mg<br>(N=XX) | dasiglucagon 0.6mg<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|
| XXXX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| XXXX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| XXXX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| XXXX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| XXXX | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | Number XXXX XXXX XXXX XXXX XXXX XXXX | Number (N=XX) XXXX xx (xx.x%) XXXX xx (xx.x%) XXXX xx (xx.x%) XXXX xx (xx.x%) XXXX xx (xx.x%) | Number (N=XX) (N=XX) XXXX xx (xx.x*) xx (xx.x*) XXXX xx (xx.x*) xx (xx.x*) XXXX xx (xx.x*) xx (xx.x*) XXXX xx (xx.x*) xx (xx.x*) XXXX xx (xx.x*) xx (xx.x*) |

Percentages are based on the total number of patients in the safety analysis set.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY RUN DATE: DDMMMYYYY hh:mm




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S

Clinical Study Report

Protocol Number: ZP4207-21052 Page x of y

# Table 14.1.3 Protocol Deviations Safety Analysis Set

| Protocol Deviations [n | dasiglucagon 0.3mg | dasiglucagon 0.6mg | Total |
|---|---|---|---|
| (%) m] | (N=XX) | (N=XX) | (N=XX) |
| Any Protocol | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Deviations[a] | | | |
| Deviation #1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Deviation #2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Deviation #3 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| etc. | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Any Major Protocol<br>Deviations[a] | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Deviation #1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Deviation #2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Deviation #3 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| etc. | xx (xx.x%) xx | xx (xx.x%) xx | xx ( xx.x%) xx |

n = Number of patients; m = Number of deviations

Percentages are based on the total number of patients in the safety analysis set. This table includes all study protocol deviations that are not COVID-19 related.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

- Only include protocol deviations that are not COVID-19 related.
- 2) Percentages are based on total number of patients in the safety set.
- 3) Include all non COVID-19 related protocol deviations in 'Any Protocol Deviations' section of the table. Include only Major non COVID-19 related protocol deviations in 'Any Major Protocol Deviations' section of the table.

RUN DATE: DDMMMYYYYY hh:mm


<sup>[</sup>a] Patients may be included in more than 1 protocol deviation category.



Zealand Pharma A/S

Protocol Number: ZP4207-21052

Page x of y

# Table 14.1.4 COVID-19 Related Protocol Deviations Safety Analysis Set

| COVID-19 Related | | dasiglucagon 0.6mg | Total |
|---|---|---|---|
| Protocol Deviations [n | dasiglucagon 0.3mg | (N=XX) | (N=XX) |
| (%) m] | (N=XX) | | |
| Any COVID-19 Related | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Protocol Deviations[2] Deviation #1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Deviation #2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Deviation #3 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| etc. | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Any Major COVID-19<br>Related Protocol<br>Deviations[a] | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Deviation #1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Deviation #2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Deviation #3 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| etc. | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |

n = Number of patients; m = Number of deviations

Percentages are based on the total number of patients in the safety analysis set.

This table includes all study protocol deviations that are COVID-19 related.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

#### Programming Note:

- 1) Only include protocol deviations that are COVID-19 related.
- 2) Percentages are based on total number of patients in the safety set.
- 3) Include all COVID-19 related protocol deviations in 'Any COVID-19 Related Protocol Deviations' section of the table. Include only Major COVID-19 related protocol deviations in 'Any Major COVID-19 Related Protocol Deviations' section of the table.

RUN DATE: DDMMMYYYY hh:mm


<sup>[</sup>a] Patients may be included in more than 1 protocol deviation category.



Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S
Clinical Study Report

Protocol Number: ZP4207-21052

Table 14.1.5 Demographic and Baseline Characteristics
Safety Analysis Set

Page x of y

| | dasiglucagon 0.3mg dasiglucagon 0.6mg | | Total |
|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) |
| age[a] (years) | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |
| ge groups | | | |
| < 2 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 2 to < 4 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| 4 to < 6 years | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| ex | | | |
| Male | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Female | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Unknown | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Undifferentiated | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Race | | | |
| American Indian or Alaska Native | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Asian | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Black or African American | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| White | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not reported | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Allowed to Ask per Local Regulation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Other | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Multiple Races Checked | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| thnicity | | | |
| Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Hispanic or Latino | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not reported | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Not Allowed to Ask per Local Regulation | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| eight (cm) | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |




| | dasiglucagon 0.3mg | dasiglucagon 0.3mg dasiglucagon 0.6mg | |
|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) |
| eight (kg) | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |
| eight groups | | | |
| < 15kg | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| >=15kg | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| MI (kg/m²) | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |
| ime Since Diabetes Diagnosis[b] (months) | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |

RUN DATE: DDMMMYYYY hh:mm

Percentages are based on the total number of patients in the safety analysis set. Height, weight and BMI obtained at Screening visit.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) This shell continues over two pages

2) Percentages are based on total number of patients in the safety set.


<sup>[</sup>a] Age on consent date

<sup>[</sup>b] Date of informed consent - date of diabetes diagnosis + 1



Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S

Clinical Study Report

Protocol Number: ZP4207-21052 Page x of y

### Table 14.1.6 Medical History Safety Analysis Set

| System Organ Class | | dasiglucagon 0.6mg | Total |
|---|---|---|---|
| Preferred term [n (%) | dasiglucagon 0.3mg | (N=XX) | (N=XX) |
| n] | (N=XX) | | |
| Any medical history | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| SOC class 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| PT Term 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| PT Term 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| ••• | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| SOC class 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| PT Term 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| PT Term 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx ( xx.x%) xx |

n = Number of patients; m = Number of events

Diabetes history not included.

Medical History terms are coded using MedDRA version 24.1. At each level of summation (SOC class, preferred name), patients reporting more than 1 event are counted only once for the patient count.

Table is sorted by descending patient count, by system organ class and preferred term.

Percentages are based on the total number of patients in the safety analysis set.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

- 1) Percentages are based on total number of patients in the safety set.
- 2) Sort by decreasing frequency of the total column by SOC and preferred term on the total column.
- 3) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table.

RUN DATE: DDMMMYYYY hh:mm

4) Please exclude any diabetes history defined as MedDDRA Preferred term =' TYPE 1 DIABETES MELLITUS'




Zealand Pharma A/S Clinical Study Report Protocol Number: ZP4207-21052

> Table 14.1.7 Prior Medications Safety Analysis Set

Page x of y

RUN DATE: DDMMMYYYY hh:mm

| ATC Class (level 2) | | dasiglucagon 0.6mg | Total |
|---|---|---|---|
| Preferred name [n (%) | dasiglucagon 0.3mg | (N=XX) | (N=XX) |
| m] | (N=XX) | | |
| Any prior medications | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| ATC Class 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred Name 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred Name 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| ••• | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| ATC Class 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred Name 1 | xx (xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred Name 2 | xx (xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| | xx (xx.x%) xx | xx (xx.x%) xx | xx (xx.x%) xx |

n = Number of patients; m = Number of occurrences

Prior medications are those that stopped before the date/time of start of study drug administration.

At each level of summation (overall, ATC class, preferred name), patients reporting more than 1 medication are counted only once for the patient count.

Table is sorted by descending patient count, by ATC level and preferred name.

Percentages are based on the total number of patients in the safety analysis set.

Terms are coded using WHODrug Global B3 format, Sep2021 release.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Percentages are based on total patient count (N).

- 2) Sort by decreasing frequency patient count, by ATC class and preferred name on the total column.
- 3) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table




Zealand Pharma A/S Clinical Study Report Protocol Number: ZP4207-21052 Page x of y

> Table 14.1.8 Concomitant Medications Safety Analysis Set

2-Jan-25

RUN DATE: DDMMMYYYYY hh:mm

| ATC Class (level 2) | | dasiglucagon 0.6mg | Total |
|---|---|---|---|
| Preferred name [n (%) | dasiglucagon 0.3mg | (N=XX) | (N=XX) |
| <u>m]</u> | (N=XX) | | |
| Any concomitant medications | xx ( xx.x%) xx | xx ( xx.x%) xx | хж ( хж.х%) хх |
| ATC Class 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred Name 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred Name 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| ••• | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| ATC Class 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred Name 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred Name 2 | xx (xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |

n = Number of patients; m = Number of occurrences

Concomitant medications are those that started, stopped or are ongoing at the date/time of start of study drug administration. At each level of summation (overall, ATC class, preferred name), patients reporting more than 1 medication are counted only once for the patient count.

Table is sorted by descending patient count, by ATC level and preferred name.

Percentages are based on the total number of patients in the safety analysis set.

Terms are coded using WHODrug Global B3 format, Sep2021 release.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Percentages are based on total patient count (N).

- 2) Sort by decreasing frequency patient count, by ATC class and preferred name on the total column.
- 3) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table




Zealand Pharma A/S

Protocol Number: ZP4207-21052

Page x of y

### Table 14.1.9 Current Diabetes Treatment Safety Analysis Set

| ATC Class (level 2) | | dasiglucagon 0.6mg | Total |
|---|---|---|---|
| Preferred name [n (%) | dasiglucagon 0.3mg | (N=XX) | (N=XX) |
| m] | (N=XX) | | |
| Any current diabetes<br>treatment | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| ATC Class 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred Name 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred Name 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| ATC Class 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred Name 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx (xx.x%) xx |
| Preferred Name 2 | xx (xx.x%) xx | xx ( xx.x%) xx | xx (xx.x%) xx |
| | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |

n = Number of patients; m = Number of occurrences

Current diabetes treatments are collected on the Diabetes Information CRF.

At each level of summation (overall, ATC class, preferred name), patients reporting more than 1 medication are counted only once for the patient count.

Table is sorted by descending patient count, by ATC level and preferred name.

Percentages are based on the total number of patients in the safety analysis set.

Terms are coded using WHODrug Global B3 format, Sep2021 release.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Percentages are based on total patient count (N).

- 2) Sort by decreasing frequency patient count, by ATC class and preferred name on the total column.
- 3) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table

RUN DATE: DDMMMYYYY hh:mm


# 14.2 Efficacy Data

# 14.2.1 Primary Efficacy Endpoint




Zealand Pharma A/S Clinical Study Report Protocol Number: ZP4207-21052

Page x of y

RUN DATE: DDMMMYYYY hh:mm

Table 14.2.1.1 Plasma Glucose Change from Baseline at 30 minutes after IMP Injection Full Analysis Set

| | dasiglucagon 0.3mg<br>(N=XX) | | _ | dasiglucagon 0.6mg<br>(N=XX) | | Total<br>(N=XX) |
|---|---|---|---|---|---|---|
| | Value | Change from baseline | Value | Change from baseline | Value | Change from<br>baseline |
| Plasma Glucose (mg/dL) at 30<br>minutes after IMP injection | | | | | | |
| n | xx | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| 95% CIs (Mean) | | (xx.x, xx.x) | | (xx.x, xx.x) | | (xx.x, xx.x) |

IMP = investigational medicinal product

Baseline is the last recorded value prior to study drug administration.

95% confidence interval for the mean plasma glucose change from baseline at 30 minutes after IMP injection, based on a t distribution. Plasma glucose change from baseline at 30 minutes after trial product injection or at the time of rescue by IV glucose. For patients who required rescue IV glucose before the time of the endpoint assessment, the last available plasma glucose taken prior to rescue IV glucose is carried forward and used for analysis.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

### Programming Note:

1) In general present mean to 1 decimal more than individual data, STD to 2 decimals more than individual data. Refer to SAP




14.2.2 Secondary Efficacy Endpoint




Zealand Pharma A/S Clinical Study Report Protocol Number: ZP4207-21052

Page x of y

RUN DATE: DDMMMYYYY hh:mm

Table 14.2.2.1 Plasma Glucose Change from Baseline at 15 minutes after IMP Injection Full Analysis Set

| | dasiglucagon 0.3mg<br>(N=XX) | | _ | dasiglucagon 0.6mg<br>(N=XX) | | Total<br>(N=XX) |
|---|---|---|---|---|---|---|
| | Value | Change from baseline | Value | Change from baseline | Value | Change from baseline |
| lasma Glucose (mg/dL) at 15 inutes after IMP injection | | | | | | |
| n | xx | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

IMP = investigational medicinal product

Baseline is the last recorded value prior to study drug administration.

Plasma glucose change from baseline at 15 minutes after trial product injection or at the time of rescue by IV glucose. For patients who required rescue IV glucose before the time of the endpoint assessment, the last available plasma glucose taken prior to rescue IV glucose is carried forward and used for analysis.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

# Programming Note:

1) In general present mean to 1 decimal more than individual data, STD to 2 decimals more than individual data. Refer to SAP




# 14.2.3 Exploratory Analysis

Zealand Pharma A/S
Protocol Number: ZP4207-21052
Page x of y

Table 14.2.3.1 Plasma Glucose Change from Baseline at 30 minutes after IMP Injection in Subjects Without Rescue IV Glucose
Full Analysis Set

#### Programming Note:

- 1) Repeat of Table 14.2.1.1 for subjects in FA but without intake of rescue INV Glucose
- 2) Remove footnote 'For patients who required rescue IV glucose before the time of the endpoint assessment, the last available plasma glucose taken prior to rescue IV glucose is carried forward and used for analysis.'

Table 14.2.3.2 Plasma Glucose Change from Baseline at 15 minutes after IMP Injection in Subjects Without Rescue IV Glucose
Full Analysis Set

#### Programming Note:

- 1) Repeat of Table 14.2.2.1 for subjects in FA but without intake of rescue INV Glucose
- 2) Remove footnote 'For patients who required rescue IV glucose before the time of the endpoint assessment, the last available plasma glucose taken prior to rescue IV glucose is carried forward and used for analysis.'




Zealand Pharma A/S Protocol Number: ZP4207-21052

Clinical Study Report Page x of y

RUN DATE: DDMMMYYYY hh:mm

2-Jan-25

Table 14.2.3.3 Plasma Glucose - untransformed and change from baseline at each time point Full Analysis Set

| | Plasma Glucose<br>(mg/dL) | _ | ngon 0.3mg<br>=XX) | | ngon 0.6mg<br>=XX) | Total<br>(N=XX) | |
|---|---|---|---|---|---|---|---|
| Time Point | | Value | Change from<br>baseline | Value | Change from<br>baseline | Value | Change from<br>baseline |
| Pre-dose | n | xx | | xx | | xx | |
| | Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| | Median | xx.x | | xx.x | | xx.x | |
| | Min, Max | xx, xx | | xx, xx | | xx, xx | |
| 15min post-dose | n | xx | xx | xx | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| 30min post-dose | n | xx | xx | xx | xx | xx | xx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

Baseline is the last recorded value prior to study drug administration.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

#### Programming Note:

1) In general present mean to 1 decimal more than individual data, STD to 2 decimals more than individual data. Refer to SAP




Zealand Pharma A/S
Protocol Number: ZP4207-21052
Page x of y

Figure 14.2.3.4 Mean glucose concentrations versus time - original scale
Full Analysis Set

| Type of Graph: | Mean concentration-time profile |
|----------------|----------------------------------------------------------|
| x-Axis | Nominal Time |
| x-Axis label | Nominal time after IMP administration (min) |
| y-Axis | Use linear scale |
| y-Axis Label | Mean plasma glucose concentration (mg/dL) |
| Additional | Same layout as figure 14.2.4.2 |
| Information | |
| Notes | Mean Line Plot per treatment |
| | Error bars showing SEM |
| | Add mean value at each plot marker rounded to 1 decimal |
| | place |
| | Add data table with number of valid cases per time point |
| Footnotes | IMP = investigational medicinal product |
| | Figure shows mean results ± SEM (Standard Error of Mean) |

# Programming Notes:

 $\ensuremath{\text{QC}}$  dataset will consist of reproducing the means and SEM plotted. So, produce a dataset with

- TRTP
- ATPTN
- Mean
- Lower bound of SEM error bar
- Upper bound of SEM error bar
- Number of valid cases

QC Dataset to be sorted by trtpn, atptn




Zealand Pharma A/S Clinical Study Report Protocol Number: ZP4207-21052

Page x of y

# Figure 14.2.3.5 Individual glucose concentrations versus time - original scale Full Analysis Set

#### Programming Note:

- This is a repeat of figure 14.2.4.3 (Spaghetti/Overlay Plot) using Plasma Glucose results. Same timepoints as used in figure 14.2.3.4

# Table 14.2.3.6 Plasma Glucose Change from Baseline at 30 minutes after IMP Injection - Sensitivity Analysis Full Analysis Set

#### Programming Note:

- This is a repeat of table 14.2.1.1 using a 2nd baseline definition with the nominal time point 'pre-dose' as baseline result

# Table 14.2.3.7 Plasma Glucose Change from Baseline at 15 minutes after IMP Injection - Sensitivity Analysis Full Analysis Set

#### Programming Note:

- This is a repeat of table 14.2.2.1 using a 2nd baseline definition with the nominal time point 'pre-dose' as baseline result

# Table 14.2.3.8 Plasma Glucose - untransformed and change from baseline at each time point- Sensitivity Analysis Full Analysis Set

#### Programming Note:

- This is a repeat of table 14.2.3.3 using a 2nd baseline definition with the nominal time point 'pre-dose' as baseline result




14.2.4 Pharmacokinetic Data




Zealand Pharma A/S Clinical Study Report Protocol Number: ZP4207-21052

Page x of y

RUN DATE: DDMMMYYYYY hh:mm

### Table 14.2.4.1 Descriptive Statistics for dasiglucagon Plasma Concentrations PK Analysis Set

Treatment Group= <dasiglucagon 0.3mg(N=XX) / dasiglucagon 0.6mg(N=XX)>

| Result (pmol/L) | Post-dose | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Pre-dose | 10min | 20min | 30min | 40min | 60min | 90min | 140min | 220min | 300min |
| n | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| CV (%) Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Max | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| Geo-Mean | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| CV (%) geom-mean[a] | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |

All concentration values below the Limit of Quantification (BLOQ) are set to zero.

Results are displayed to 3 significant digits.

[a] Geometric mean CV (%) is calculated as  $[\exp(SD^2)-1]^{1/2}*100$ , where SD is standard deviation of the natural-log transformed data.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

- 1) In general present mean to 1 decimal more than individual data, STD to 2 decimals more than individual data. Refer to SAP
- 2) For post-dose samples, the planned sampling time will be used in summary tables.
- 3) For all pre-dose samples, the sampling time will be set to zero.
- 4) All concentration values below the Limit of Quantification (BLOQ) will be set to zero.
- 5) Missing post-dose values will not be replaced
- 6) See further details in the SAP
- 7) Table will be created for each treatment group




 ZP4207-21052
 2-Jan-25

 Zealand Pharma A/S
 Clinical Study Report

 Protocol Number: ZP4207-21052
 Page x of y

Figure 14.2.4.2 Mean dasiglucagon Concentration-time Profile - linear scale

PK Analysis Set

| Type of Graph: | Mean concentration-time profile |
|----------------|----------------------------------------------------------|
| x-Axis | See mock on next page |
| x-Axis label | Nominal time after IMP administration (min) |
| y-Axis | Use linear scale |
| | Use same scaling of y axis for all patients |
| y-Axis Label | Mean dasiglucagon concentration (pmol/L) |
| Additional | See next page for mock. |
| Information | |
| Notes | Mean Line Plot |
| | Error bars showing SEM |
| | Add data table as in example plot |
| Footnotes | IMP = investigational medicinal product |
| | Figure shows mean results ± SEM (Standard Error of Mean) |
| | Results BLQ are set to 0 pmol/L |

# Programming Notes:

 $\ensuremath{\text{QC}}$  dataset will consist of reproducing the means and SEM plotted. So, produce a dataset with

- TRTP
- ATPTN
- Mean
- Lower bound of SEM error bar
- Upper bound of SEM error bar
- Number of valid cases

QC Dataset to be sorted by trtpn, atptn




Zealand Pharma A/S
Protocol Number: ZP4207-21052
Page x of y



 $\label{eq:IMP} \begin{tabular}{ll} IMP = investigational medicinal product\\ Figure shows mean results <math>\pm$  SEM (Standard Error of Mean)\\ Results BLQ are set to 0 pmol/L \\ \end{tabular}




Zealand Pharma A/S

Clinical Study Report Protocol Number: ZP4207-21052

> Figure 14.2.4.3 Mean dasiglucagon Concentration-time Profile - semi-log scale PK Analysis Set

| Type of Graph: | Mean concentration-time profile |
|----------------|----------------------------------------------------------|
| x-Axis | See mock on next page |
| x-Axis label | Nominal time after IMP administration (min) |
| y-Axis | Use semi-log scale |
| | Use same scaling of y axis for all patients |
| y-Axis Label | Mean dasiglucagon concentration (pmol/L) |
| Additional | |
| Information | |
| Notes | Mean Line Plot |
| | Error bars showing SEM |
| | Add data table as in example plot |
| Footnotes | IMP = investigational medicinal product |
| | Figure shows mean results ± SEM (Standard Error of Mean) |
| | Results BLQ are set to 0 pmol/L |

## Programming Note:

1) Repeat of Figure 14.2.4.2 on Semi-log scale

QC dataset will consist of reproducing the means and SEM plotted. So, produce a dataset with

- TRTP
- ATPTN
- Mean
- Lower bound of SEM error bar
- Upper bound of SEM error bar
- Number of valid cases

QC Dataset to be sorted by trtpn, atptn Zealand Pharma A/S Clinical Study Report

Protocol Number: ZP4207-21052

CONFIDENTIAL Page 62/152 Page x of y

Page x of y



Figure 14.2.4.4 Individual overlayed dasiglucagon Concentration-time Profiles - linear scale PK Analysis Set

| Type of Graph: | Spaghetti plots |
|---|---|
| x-Axis | See mock on next page |
| x-Axis label | Actual time after IMP administration (min) |
| y-Axis | Use linear scale |
| | Use same scaling of y axis for all patients |
| y-Axis Label | dasiglucagon concentration (pmol/L) |
| Additional | See next page for mock. |
| Information | |
| Notes | Spaghetti Plot, one plot per dose |
| | Use different color (red/blue as in previous plot) for the 2 |
| | dose groups |
| Footnotes | IMP = investigational medicinal product |
| | For individual concentration-time profiles, the actual |
| | sampling times is used. |

# Programming Notes:

QC dataset will consist of reproducing the results plotted. So, produce a dataset with

- TRTP
- SUBJID
- ARELIM2
- AVAL

QC Dataset to be sorted by trtpn, subjid, areltm2




Sample Plot (from other study)

Zealand Pharma A/S Clinical Study Report

Protocol Number: ZP4207-17086 Page 1 of 2

14.4.1.5 Figure: Individual analyte concentrations versus time curves - original scale, FAS

Treatment=dasiglucagon






Clinical Study Report Zealand Pharma A/S Protocol Number: ZP4207-21052

> Figure 14.2.4.5 Individual dasiglucagon Concentration-time Profiles - linear scale PK Analysis Set

2-Jan-25

Page x of y

| Type of Graph: | Individual Patient concentration-time profiles |
|----------------|--------------------------------------------------------|
| x-Axis | See mock on next page |
| x-Axis label | Actual time after IMP administration (min) |
| y-Axis | Use linear scale |
| | Use same scaling of y axis for all patients |
| y-Axis Label | dasiglucagon concentration (pmol/L) |
| Additional | See next page for mock. |
| Information | |
| Notes | Panel Plot, separate panel for each dosing group |
| Footnotes | IMP = investigational medicinal product |
| | For individual concentration-time profiles, the actual |
| | sampling times is used. |

# Programming Notes:

QC dataset will consist of reproducing the results plotted. So, produce a dataset with

- TRTP
- SUBJID
- ARELIM2
- AVAL

QC Dataset to be sorted by trtpn, subjid, areltm2

CONFIDENTIAL Page 65/152 Zealand Pharma A/S ZP4207-21052

Treatment=< dasiglucagon 0.6mg/ dasiglucagon 0.6mg >






Clinical Study Report Zealand Pharma A/S Protocol Number: ZP4207-21052 Page x of y

Figure 14.2.4.6 Individual dasiglucagon Concentration-time Profiles - Semi-log scale PK Analysis Set

2-Jan-25

| Type of Graph: | Individual Patient concentration-time profiles |
|----------------|--------------------------------------------------------|
| x-Axis | See mock. |
| x-Axis label | Actual time after IMP administration (min) |
| y-Axis | Use semi-log scale |
| | Use same scaling of y axis for all patients |
| y-Axis Label | dasiglucagon concentration (pmol/L) |
| Additional | |
| Information | |
| Notes | Panel Plot, separate panel for each dosing group |
| Footnotes | IMP = investigational medicinal product |
| | For individual concentration-time profiles, the actual |
| | sampling times is used. |

# Programming Note:

2) Repeat of Figure 14.2.4.5 on Semi-log scale

# Programming Notes:

QC dataset will consist of reproducing the results plotted. So, produce a dataset with

- TRTP
- SUBJID
- ARELTM2
- AVAL

QC Dataset to be sorted by trtpn, subjid, areltm2




Zealand Pharma A/S Protocol Number: ZP4207-21052

Clinical Study Report Page x of y

RUN DATE: DDMMMYYYY hh:mm

2-Jan-25

### Table 14.2.4.7 Descriptive Statistics for PK Parameters PK Analysis Set

Treatment Group= <dasiglucagon 0.3mg(N=XX)/ dasiglucagon 0.6mg(N=XX)>

| Statistic | Cmax<br>(pmol/L) | Tmax<br>(h) | Lambda z<br>(1/h) | T1/2<br>(h) | AUC<br>(0-<br>30mins)<br>(unit) | AUC<br>(0-300)<br>(unit) | AUC<br>(0-tlast)<br>(unit) | AUC<br>(0-inf)<br>(unit) | CL/f<br>(unit) | Vz/f<br>(unit) | MRT<br>(unit) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| n | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Mean (SD) | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) | (xx.xx) |
| Mean CV (%) | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Geometric Mean | xx, xx | - | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Geometric Mean CV (%) [a] | xx.x | - | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |

Results are displayed to 3 significant digits.

[a] Geometric CV (%) is calculated as  $[\exp(SD^2)-1]^{1/2}*100$ , where SD is standard deviation of the natural-log transformed data.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

- 1) Extend to a 2<sup>nd</sup> page if not sufficient space to display full length of numbers
- 2) Order PK parameters per the order in Section 12.1 of the SAP.
- 3) The geometric mean and CV% for the geometric mean will not be calculated for  $T_{max}$


14.3 Safety Data

14.3.1 Adverse Events




Zealand Pharma A/S Protocol Number: ZP4207-21052

Clinical Study Report Page x of y

RUN DATE: DDMMMYYYY hh:mm

2-Jan-25

# Table 14.3.1.1 Overall Summary of Adverse Events Safety Analysis Set

| Adverse Event Category [n (%) m] | dasiglucagon 0.3mg<br>(N=XX) | dasiglucagon 0.6mg<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|
| AEs that occurred during screening | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Treatment-emergent adverse events (TEAEs) | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Treatment-emergent adverse events (TEAEs) occurring within 12 hours after dosing | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| TEAEs of special interest | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| TEAEs which are other important events | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| TEAEs which are injection site reactions[a] | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| TEAEs which are related[b] to the study drug | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Serious TEAEs | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Serious TEAEs which are related to the study drug | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Adverse events leading to death | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |

n = Number of patients; m = Number of occurrences

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY


<sup>[</sup>a] Based on investigator assessment on the eCRF

<sup>[</sup>b] Probable and possible relationships are included under the category related. In case of missing relationship will be set to related for the analysis.

Patients reporting more than 1 event are counted only once for the patient count.

Percentages are based on the total number of patients in the safety analysis set for the given dose group.

Treatment-emergence is defined as those AEs that occurred after dosing and those existing AEs that worsened during the study.



Zealand Pharma A/S Clinical Study Report Protocol Number: ZP4207-21052

Page x of y

Table 14.3.1.2 Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Safety Analysis Set

| ystem organ class<br>Preferred term [n (%) m] | dasiglucagon 0.3mg<br>(N=XX) | dasiglucagon 0.6mg<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|
| ny treatment-emergent adverse events | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| ystem organ class 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred term 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred term 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred term 3 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| ystem organ class 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred term 1 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |
| Preferred term 2 | xx ( xx.x%) xx | xx ( xx.x%) xx | xx ( xx.x%) xx |

n = Number of patients; m = Number of events

Adverse events are coded using MedDRA version 24.1. At each level of summation (system organ class, preferred term) patients reporting more than 1 event are included only once.

Table is sorted by descending patient count, by system organ class and preferred term.

Percentages are based on the total number of patients in the safety analysis set for the given dose group.

Treatment-emergence is defined as those AEs that occurred after dosing and those existing AEs that worsened during the study.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

# Programming Note:

- 1) Percentages are based on total subject count (N) for each column
- 2) Sort by decreasing frequency of patients, by SOC and preferred term on the total column.
- 3) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table




Zealand Pharma A/S

ZP4207-21052

Zealand Pharma A/S

Clinical Study Report

Protocol Number: ZP4207-21052 Page x of y

# Table 14.3.1.3 Treatment-Emergent Adverse Events occurring within 12 hours after dosing by System Organ Class and Preferred Term Safety Analysis Set

n = Number of patients; m = Number of events

Adverse events are coded using MedDRA version 24.1. At each level of summation (system organ class, preferred term) patients reporting more than 1 event are included only once.

Table is sorted by descending patient count, by system organ class and preferred term.

Percentages are based on the total number of patients in the safety analysis set for the given dose group.

Treatment-emergence is defined as those AEs that occurred after dosing and those existing AEs that worsened during the study.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

#### Programming Note:

- 1) Repeat of table 14.3.1.2 for treatment-emergent adverse events that occurred within 12 hours after dosing only.
- 2) Percentages are based on total subject count (N) for each column
- 3) Sort by decreasing frequency of patients, by SOC and preferred term on the total column.
- 4) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table



Protocol Number: ZP4207-21052

## Table 14.3.1.4 Adverse Events that occurred during Screening, by System Organ Class and Preferred Term Safety Analysis Set

n = Number of patients; m = Number of events

Adverse events are coded using MedDRA version 24.1. At each level of summation (system organ class, preferred term) patients reporting more than 1 event are included only once.

Table is sorted by descending patient count, by system organ class and preferred term.

Percentages are based on the total number of patients in the safety analysis set for the given dose group.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

Page x of y

#### Programming Note:

- 5) Repeat of table 14.3.1.2 for adverse events that occurred during screening only.
- 6) Percentages are based on total subject count (N) for each column
- 7) Sort by decreasing frequency of patients, by SOC and preferred term on the total column.
- 8) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table
- 9) Set first row in table to 'Any adverse events' instead of 'Any treatment-emergent adverse events'.




Protocol Number: ZP4207-21052

## Table 14.3.1.5 Treatment-Emergent Adverse Events of Special Interest, by System Organ Class and Preferred Term Safety Analysis Set

n = Number of patients; m = Number of events

Adverse events are coded using MedDRA version 24.1. At each level of summation (system organ class, preferred term) patients reporting more than 1 event are included only once.

Table is sorted by descending patient count, by system organ class and preferred term.

Percentages are based on the total number of patients in the safety analysis set for the given dose group.

Treatment-emergence is defined as those AEs that occurred after dosing and those existing AEs that worsened during the study.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

Page x of y

- Programming Note:
  - 1) Repeat of table 14.3.1.2 for treatment-emergent adverse events of special interest only.
  - 2) Percentages are based on total subject count (N) for each column
  - 3) Sort by decreasing frequency of patients, by SOC and preferred term on the total column.
  - 4) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table




Protocol Number: ZP4207-21052 Page x of y

# Table 14.3.1.6 Treatment-Emergent Adverse Events that are Other Important Events, by System Organ Class and Preferred Term Safety Analysis Set

n = Number of patients; m = Number of events

Adverse events are coded using MedDRA version 24.1. At each level of summation (system organ class, preferred term) patients reporting more than 1 event are included only once.

Table is sorted by descending patient count, by system organ class and preferred term.

Percentages are based on the total number of patients in the safety analysis set for the given dose group.

Treatment-emergence is defined as those AEs that occurred after dosing and those existing AEs that worsened during the study.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY Programming Note:

RUN DATE: DDMMMYYYY hh:mm

- 1) Repeat of table 14.3.1.2 for treatment-emergent adverse events that are other important events only.
  2) Percentages are based on total subject count (N) for each column
- 3) Sort by decreasing frequency of patients, by SOC and preferred term on the total column.
- 4) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table




Zealand Pharma A/S

ZP4207-21052

Zealand Pharma A/S

Clinical Study Report

Protocol Number: ZP4207-21052

Table 14.3.1.7 Treatment-Emergent Adverse Events that are Injection Site Reactions, by System Organ Class and Preferred Term
Safety Analysis Set

n = Number of patients; m = Number of events

Adverse events are coded using MedDRA version 24.1. At each level of summation (system organ class, preferred term) patients reporting more than 1 event are included only once.

Table is sorted by descending patient count, by system organ class and preferred term.

Percentages are based on the total number of patients in the safety analysis set for the given dose group.

Treatment-emergence is defined as those AEs that occurred after dosing and those existing AEs that worsened during the study.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY Programming Note:

RUN DATE: DDMMMYYYYY hh:mm

Page x of y

- Repeat of table 14.3.1.2 for treatment-emergent adverse events that are injection site reactions.
   Percentages are based on total subject count (N) for each column
  - 3) Sort by decreasing frequency of patients, by SOC and preferred term on the total column.
  - 4) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S

Clinical Study Report

Protocol Number: ZP4207-21052

## Table 14.3.1.8 Treatment-Emergent Adverse Events that are IMP Related, by System Organ Class and Preferred Term Safety Analysis Set

n = Number of patients; m = Number of events; IMP = investigational medicinal product

IMP related: Adverse events which were assessed by the investigator with a reported relationship to IMP of 'Possible' or 'Probable'. Adverse events are coded using MedDRA version 24.1. At each level of summation (system organ class, preferred term) patients reporting more than 1 event are included only once.

Table is sorted by descending patient count, by system organ class and preferred term.

Percentages are based on the total number of patients in the safety analysis set for the given dose group.

Treatment-emergence is defined as those AEs that occurred after dosing and those existing AEs that worsened during the study.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYYY hh:mm

Page x of y

Programming Note:

- 1) Repeat of table 14.3.1.2 for treatment-emergent adverse events with a reported relationship to study treatment of 'Possible' or 'Probable'.
- 2) Percentages are based on total subject count (N) for each column
- 3) Sort by decreasing frequency of patients, by SOC and preferred term on the total column.
- 4) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table




Zealand Pharma A/S Clinical
Protocol Number: ZP4207-21052

Page x of y

## Table 14.3.1.9 Serious Treatment-Emergent Adverse Events, by System Organ Class and Preferred Term Safety Analysis Set

n = Number of patients; m = Number of events

Adverse events are coded using MedDRA version 24.1. At each level of summation (system organ class, preferred term) patients reporting more than 1 event are included only once.

Table is sorted by descending patient count, by system organ class and preferred term.

Percentages are based on the total number of patients in the safety analysis set for the given dose group.

Treatment-emergence is defined as those AEs that occurred after dosing and those existing AEs that worsened during the study.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY Programming Note:

RUN DATE: DDMMMYYYY hh:mm

- 1) Repeat of table 14.3.1.2 for serious treatment-emergent adverse events.
- 2) Percentages are based on total subject count (N) for each column
- 3) Sort by decreasing frequency of patients, by SOC and preferred term on the total column.
- 4) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table
- 5) Set first row in table to 'Any serious treatment-emergent adverse events' instead of 'Any treatment-emergent adverse events'.

61




Zealand Pharma A/S

ZP4207-21052

Zealand Pharma A/S

Clinical Study Report

Protocol Number: ZP4207-21052 Page x of y

## Table 14.3.1.10 Serious Treatment-Emergent Adverse Events that are IMP Related, by System Organ Class and Preferred Term Safety Analysis Set

n = Number of patients; m = Number of events; IMP = investigational medicinal product

IMP related: Adverse events which were assessed by the investigator with a reported relationship to IMP of 'Possible' or 'Probable'. Adverse events are coded using MedDRA version 24.1. At each level of summation (system organ class, preferred term) patients reporting more than 1 event are included only once.

Table is sorted by descending patient count, by system organ class and preferred term.

Percentages are based on the total number of patients in the safety analysis set for the given dose group.

Treatment-emergence is defined as those AEs that occurred after dosing and those existing AEs that worsened during the study.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

Programming Note:

- 1) Repeat of table 14.3.1.2 for serious treatment-emergent adverse events with a reported relationship to study treatment of 'Possible' or 'Probable'.
- 2) Percentages are based on total subject count (N) for each column
- 3) Sort by decreasing frequency of patients, by SOC and preferred term on the total column.
- 4) Any uncoded terms to be displayed under a SOC 'Uncoded' and then the verbatim term for the PT (in all capital letters) and to be sorted to appear at the bottom of the table




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 Zealand Pharma A/S

Protocol Number: ZP4207-21052

2-Jan-25 Clinical Study Report Page x of y

## Table 14.3.1.11 Local Tolerability Assessment Safety Analysis Set

| .6mg(N=XX)>Time point | Type of Reaction | Mild | Moderate | Severe | Total |
|---|---|---|---|---|---|
| osing: 30 minutes post dose | Spontaneous Pain | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Pain On Palpation | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Itching | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Redness | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Edema | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Induration/Infiltration | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Other | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| osing: 120 minutes post dose | Spontaneous Pain | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Pain On Palpation | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Itching | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Redness | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Edema | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Induration/Infiltration | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Other | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| osing: 300 minutes post dose | Spontaneous Pain | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Pain On Palpation | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Itching | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Redness | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Edema | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Induration/Infiltration | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Other | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| ollow-up | Spontaneous Pain | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Pain On Palpation | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Itching | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Redness | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Edema | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Induration/Infiltration | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | Other | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

RUN DATE: DDMMMYYYY hh:mm

Percentages are based on the number of patients who had a local tolerability assessment at that timepoint.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Only display 'Other' rows where there are counts populated.




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052
2-Jan-25

14.3.2 Listings of Deaths, Other Serious and Significant Adverse Events




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052

2-Jan-25 Clinical Study Report Zealand Pharma A/S Page x of y Protocol Number: ZP4207-21052

## Listing 14.3.2.1 Serious Adverse Events Safety Analysis Set

| Treatment<br>nt<br>Group | | | System Organ<br>Class/ | Start Date Time<br>(Study Day[b])/ | | Action<br>Taken<br>with | | AESI <sup>[c]</sup> / | | | Plasma | Glucose |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patien | t AE | | Preferred Term/<br>Verbatim Term | End Date Time<br>(Study Day <sup>[b]</sup> ) | Severity/<br>Causality | Study | Outcome | - | tType of Other<br>Important Event <sup>[d]</sup> | | .Start<br>Time Source | Value<br>(unit) |
| xxxx | xx | Y/<br>N | xxxx/<br>xxxx/<br>xxxx | YYYY-MM-DDTHH:MM<br>(Day XX)/<br>YYYY-MM-DDTHH:MM<br>(Day XX) | Possible | Dose<br>Reduced | Unknown | N/<br>Y | Infection/ Overdose/ Abuse or misuse/ Error/ Accidental exposure/ Risk of liver injury | Y | HH:MM xxxxx | xxx<br>(xxx) |
| | | | | YYYY-MM-DD<br>(Day XX)/<br>UNKNOWN | | | | | | | | |

Programming note:

1) This shell continues over two pages




Zealand Pharma A/S
Statistical Analysis Plan
ZP4207-21052
2-Jan-25

Zealand Pharma A/S

Protocol Number: ZP4207-21052

Clinical Study Report
Page x of y

RUN DATE: DDMMMYYYY hh:mm

#### Listing 14.3.2.1 Serious Adverse Events Safety Analysis Set

| | | | | | | Ser | ious Criteria Met | | |
|---|---|---|---|---|---|---|---|---|---|
| | | System Organ | Start Date Time | | | | Hospitalization | | |
| Treatment | | Class/ | (Study Day[b])/ | Congenital | | | or Prolongation | | Other Serious |
| Group - | AE TE- | Preferred Term/ | End Date | Anomaly or | Significan | t | of | Life | Important |
| Patient ID | # AE[a] | Verbatim Term | (Study Day <sup>[b]</sup> ) | Birth Defect | Disability | Death | Hospitalization | Threatening | Medical Event |
| xxxx | xx Y/ | xxxx/ | YYYY-MM-DDTHH:MM | Y/N | Y/N | Y/N | Y/N | Y/N | Y:xxxxxx |
| | N | xxxx/ | (XX) / | | | | | | |
| | | xxxx | YYYY-MM-DD | | | | | | |
| | | | (XX) | | | | | | |
| | | | YYYY-MM-DD | | | | | | |
| | | | (XX) / | | | | | | |
| | | | ONGOING | | | | | | |

[d] Infection=Suspicion of transmission of infectious agents via the trial product; Overdose=Overdose of the trial product; Abuse or misuse=Suspected abuse or misuse of the trial product; Error=Medication error involving the trial product; Accidental exposure=Inadvertent or accidental exposure to the trial product; Risk of liver injury=Risk of liver injury defined as ALT or AST > 3 x ULN and total bilirubin > 2 x ULN, where no alternative etiology exists;

[e] Hypoglycemia Episode?

Adverse events are coded using MedDRA version 24.1.

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

#### Programming note:

- 1) This shell continues over two pages
- 2) Sort by patient, start date and end date.


<sup>[</sup>a] TEAE: Treatment-emergent AE

<sup>[</sup>b] Study day is derived relative to the date/time of start of study drug administration.

<sup>[</sup>c] AESI: AE of special interest



Protocol Number: ZP4207-21052

Page x of y

#### Listing 14.3.2.2 Adverse Events Leading to Death Safety Analysis Set

[a] TEAE: Treatment-emergent AE

- [b] Study day is derived relative to the date/time of start of study drug administration.
- [c] AESI: AE of special interest
- [d] Infection=Suspicion of transmission of infectious agents via the trial product; Overdose=Overdose of the trial product; Abuse or misuse=Suspected abuse or misuse of the trial product; Error=Medication error involving the trial product; Accidental exposure=Inadvertent or accidental exposure to the trial product; Risk of liver injury=Risk of liver injury defined as ALT or AST > 3 x ULN and total bilirubin > 2 x ULN, where no alternative etiology exists;

RUN DATE: DDMMMYYYY hh:mm

[e] Hypoglycemia Episode?

Adverse events were coded using MedDRA version 24.1.

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

- 1) Repeat Listing 14.3.2.1 for records where 'Outcome' = 'Fatal'.
- 2) Sort by patient, start date and end date.




Protocol Number: ZP4207-21052

## 14.3.3 Narratives of Deaths, Other Serious and Certain Other Significant Adverse Events

Page x of y

Please refer to section 12.3.2 of the CSR

PROGRAM SOURCE: tlf-###, DATA CUT-OFF DATE: DDMMMYYYY RUN DATE: DDMMMYYYY hh:mm

Programming Note: Create an empty table using the %nodata macro with that reference as message




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

14.3.4 Abnormal Laboratory Value Listing (Each Patient)




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
2-Jan-25

 ZP4207-21052
 2-Jan-25

 Zealand Pharma A/S
 Clinical Study Report

 Protocol Number: ZP4207-21052
 Page x of y

Listing 14.3.4.1 Abnormal Laboratory Values
Safety Analysis Set

| Treatment<br>Group - | | | | | | Change<br>from | Normal |
|---|---|---|---|---|---|---|---|
| Patient ID | Category | Parameter (unit) | Visit[a] | Date/Time of Collection (Study Day[b]) | Result[c] | Baseline | Range |
| xxxx | Hematology | xxxx | Screening (BL)<br>Follow-up | YYYY-MM-DDTHH:MM (Day XX)<br>YYYY-MM-DDTHH:MM (Day XX) | xxxx (L) | xxxx | xx-xx |
| | | xxxx | Screening | | | | |

RUN DATE: DDMMMYYYY hh:mm

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

### Programming Note:

- 1) Only display Abnormal lab results (i.e. where the result does not fall within the normal range)
- 2) Sort by Patient, category (Hematology, chemistry, then coagulation), parameter and date/time
- 3) After each parameter add a blank line


<sup>[</sup>a] BL: Baseline Flag

<sup>[</sup>b] Study day is derived relative to the date/time of start of study drug administration.

<sup>[</sup>c] L: Below Normal Range, H: Above Normal Range



Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

14.3.5 Extent of Exposure




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S
Clinical Study Report

Protocol Number: ZP4207-21052

Page x of y

## Table 14.3.5.1 Hypoglycemia Induction Procedure Safety Analysis Set

| | dasiglucagon 0.3mg<br>(N=XX) | dasiglucagon 0.6mg<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|
| Typoglycemia induction procedure performed? | | | |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| MDI User: Duration between last basal dose before the hypoglycemia procedure and time when hypoglycemia procedure was initiated (min) | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Pump User: Duration between stop of insulin pump and ime when hypoglycemia procedure was initiated (min) | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |
| otal amount of insulin administered to induce hypoglycemia (IU) | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |
| clucose administered intravenously prior to dosing? | | | |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| otal amount of glucose administered (mL) | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |




## Zealand Pharma A/S ZP4207-21052

Statistical Analysis Plan 2-Jan-25

| | dasiglucagon 0.3mg<br>(N=XX) | dasiglucagon 0.6mg<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|
| Rescue IV Glucose given after dosing? | | | |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Fime to first IV glucose infusion (min) | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |

Time to first IV glucose infusion (min): Time of start of first glucose administration - Time of administration of study medication.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY hh:mm




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

14.3.6 Other Safety Data




Protocol Number: ZP4207-21052

Figure 14.3.6.1 Continuous Glucose Monitoring - Individual Glucose Concentration-time Profiles
Safety Analysis Set

Page x of y

| Type of Graph: | Individual Patient concentration-time profiles |
|---|---|
| x-Axis | Actual time from the time of stopping patient's insulin pump (h) |
| x-Axis label | Actual time from the time of stopping patient's insulin pump (h) |
| y-Axis | Use linear scale Use same scaling of y axis for all patients |
| y-Axis Label | Glucose concentration (mg/dL) Secondary y axis: mmol/L Results are converted into the unit 'mmol/L' by using the conversion factor 0.0555 (i.e. Glucose [mmol/L]=Glucose [mg/dL] *0.0555). |
| Additional<br>Information | See next page for mock. |
| Notes | Panel Plot, separate panel for each dosing group. One page per subject. |
| Footnotes | Glucose-time profiles based on continuous glucose monitoring from the time of stopping the patient's insulin pump to 300 minutes after dasiglucagon administration. |

#### Programming Notes:

 $\ensuremath{\textit{QC}}$  dataset will consist of reproducing the results plotted. So, produce a dataset with

- TRTP
- USUBJID
- ARELIM
- AVAL (where PARAMCD=GLUCMG)
- AVAL (where PARAMCD=GLUCMOL)

QC Dataset to be sorted by trtpn, usubjid, areltm




Treatment=dasiglucagon 0.3mg






 Zealand Pharma A/S
 Statistical Analysis Plan

 ZP4207-21052
 2-Jan-25

 Zealand Pharma A/S
 Clinical Study Report

Protocol Number: ZP4207-21052

Figure 14.3.6.2 Glucose Analyser Data- Individual Glucose Concentration-time Profiles
Safety Analysis Set

Page x of y

| Type of Graph: | Individual Patient concentration-time profiles |
|---|---|
| x-Axis | Relative time from start of first dosing of IMP |
| x-Axis label | Actual time from the time of first dosing (min) |
| y-Axis | Use linear scale Use same scaling of y axis for all patients |
| y-Axis Label | Glucose Analyser concentration (mg/dL) |
| Additional<br>Information | Similar layout as plot as figure 14.3.6.1 using Glucose analyser data and only one y-axis |
| Notes | Panel Plot, separate panel for each dosing group |
| Footnotes | Glucose-time profiles based on Glucose Analyser Data. |

## Programming Notes:

QC dataset will consist of reproducing the results plotted. So, produce a dataset with

- TRTP
- USUBJID
- ARELIM
- AVAL

QC Dataset to be sorted by trtpn, usubjid, areltm


Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052
2-Jan-25

17.1.1.1 14.3.6.3 Laboratory Data




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S

Clinical Study Report

Protocol Number: ZP4207-21052

## Table 14.3.6.3.1 Hematology Results Safety Analysis Set

Page x of y

RUN DATE: DDMMMYYYY hh:mm

| | _ | agon 0.3mg<br>=XX) | _ | ngon 0.6mg<br>=XX) | | tal<br>=XX) |
|---|---|---|---|---|---|---|
| Lab parameter (unit) | | Change from | | Change from | | Change from |
| Time point | Value | baseline | Value | baseline | Value | baseline |
| Lab parameter (unit) | | | | | | |
| Baseline | | | | | | |
| n | xx | | xx | | xx | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | xx.x | | xx.x | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | |
| Follow-up | | | | | | |
| n | xx | xx | xx | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

Baseline is the last assessment prior to study drug administration.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

2) In general present mean to 1 decimal more than individual data, STD to 2 decimals more than individual data. Refer to SAP

3) Order parameters alphabetically




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 2-Jan-25

Clinical Study Report Zealand Pharma A/S Protocol Number: ZP4207-21052

> Table 14.3.6.3.2 Hematology Results - Reference Range Analysis Safety Analysis Set

Page x of y

RUN DATE: DDMMMYYYY hh:mm

| Lab parameter (unit)<br>Time point | dasiglucagon 0.3mg<br>(N=XX) | dasiglucagon 0.6mg<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|
| Lab parameter (unit) | | | |
| Baseline | | | |
| Low | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Normal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| High | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Follow-up | | | |
| Low | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Normal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| High | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Baseline is the last assessment prior to study drug administration.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Summarize the counts and percentages of the results above/below/within the reference range, for each parameter at each visit.




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S

Clinical Study Report

Zealand Pharma A/S Clini Protocol Number: ZP4207-21052

Page x of y

RUN DATE: DDMMMYYYY hh:mm

## Table 14.3.6.3.3 Chemistry Results Safety Analysis Set

Baseline is the last assessment prior to study drug administration. Results reported as below the detection limit are set to missing in this table.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

3) Repeat of Table 14.3.6.3.1 for Chemistry parameters

4) In general present mean to 1 decimal more than individual data, STD to 2 decimals more than individual data. Refer to SAP

5) Order parameters alphabetically




Protocol Number: ZP4207-21052

# Table 14.3.6.3.4 Chemistry Results - Reference Range Analysis Safety Analysis Set

Baseline is the last assessment prior to study drug administration.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

Page x of y

#### Programming Note:

- 1) Repeat of Table 14.3.6.3.2 for Chemistry parameters
- 2) Summarize the counts and percentages of the results above/below/within the reference range, for each parameter at each visit.




Protocol Number: ZP4207-21052

## Table 14.3.6.3.5 Coagulation Results Safety Analysis Set

Page x of y

Baseline is the last assessment prior to study drug administration.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY hh:mm

## Programming Note:

- 1) Repeat of Table 14.3.6.3.1 for Chemistry parameters
- 2) In general present mean to 1 decimal more than individual data, STD to 2 decimals more than individual data. Refer to SAP
- 3) Order parameters alphabetically




Protocol Number: ZP4207-21052

# Table 14.3.6.3.6 Coagulation Results - Reference Range Analysis Safety Analysis Set

Baseline is the last assessment prior to study drug administration.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

Page x of y

#### Programming Note:

- 1) Repeat of Table 14.3.6.3.3 for Chemistry parameters
- 2) Summarize the counts and percentages of the results above/below/within the reference range, for each parameter at each visit.




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
2-Jan-25

Zealand Pharma A/S
Protocol Number: ZP4207-21052
Page x of y

## Table 14.3.6.3.7 Immunogenicity Safety Analysis Set

| | dasiglucagon 0.3mg<br>(N=XX) | dasiglucagon 0.6mg<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|
| | , | , | • |
| Occurrence of ADA | | | |
| No | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Yes | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Missing | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Overall ADA including treatment-induced ADA and treatment-boosted ADA.

Percentages is derived from patients having an ADA assessment.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY hh:mm




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S
Clinical Study Report

Protocol Number: ZP4207-21052

Page x of y

## Table 14.3.6.4 Vital Signs Safety Analysis Set

| | | ngon 0.3mg<br>=XX) | | gon 0.6mg<br>XX) | | tal<br>-XX) |
|---|---|---|---|---|---|---|
| Vital signs parameter (unit)<br>Time point | Value | Change from baseline | Value | Change from baseline | Value | Change from |
| Time point | Varue | Dubollio | Value | Dubolino | varuo | Dubelline |
| /ital signs parameter (unit) | | | | | | |
| Screening | | | | | | |
| n | xx | | xx | | xx | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | xx.x | | xx.x | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | |
| Baseline | | | | | | |
| n | xx | | xx | | xx | |
| Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| Median | xx.x | | xx.x | | xx.x | |
| Min, Max | xx, xx | | xx, xx | | xx, xx | |
| Dosing: 30 minutes post- | | | | | | |
| lose | | | | | | |
| | xx | xx | xx | xx | xx | xx |
| n | ** | | | | | |
| n<br>Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| | | xx.x (xx.xx)<br>xx.x | xx.x (xx.xx)<br>xx.x | xx.x (xx.xx)<br>xx.x | xx.x (xx.xx)<br>xx.x | xx.x (xx.xx<br>xx.x |
| Mean (SD) | xx.x (xx.xx) | , , | , , | | | - |
| Mean (SD)<br>Median | xx.x (xx.xx)<br>xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Mean (SD)<br>Median<br>Min, Max | xx.x (xx.xx)<br>xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Mean (SD)<br>Median<br>Min, Max | xx.x (xx.xx)<br>xx.x | xx.x | xx.x | xx.x | xx.x | xx.x |
| Mean (SD) Median Min, Max nterpretation Baseline Normal | xx.x (xx.xx)<br>xx.x<br>xx, xx | xx.x<br>xx, xx<br>xx ( xx.x%) | xx.x<br>xx, xx<br>xx ( xx.x%) | xx.x<br>xx, xx<br>xx ( xx.x%) | xx.x<br>xx, xx<br>xx ( xx.x%) | xx.x<br>xx, xx<br>xx ( xx.x% |
| Mean (SD) Median Min, Max nterpretation Baseline | xx.x (xx.xx)<br>xx.x<br>xx, xx | xx.x<br>xx, xx | xx.x<br>xx, xx | xx.x<br>xx, xx | xx.x<br>xx, xx | xx.x<br>xx, xx |

Baseline is the last assessment prior to study drug administration.




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

Percentages are based on the total number of patients in the safety analysis set.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

## Programming Note:

- 1) In general present mean to 1 decimal more than individual data, STD to 2 decimals more than individual data.
- 2) Order parameters as follows: Height, Weight, BMI, Temperature, Systolic BP, Diastolic BP, Fulse, Interpretation.
- 3) Continue for each parameter at screening, baseline and each post-baseline assessment
- 4) Start a new page after each parameter




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
2-Jan-25

Zealand Pharma A/S Protocol Number: ZP4207-21052 Clinical Study Report
Page x of y

RUN DATE: DDMMMYYYY hh:mm

## Table 14.3.6.5 ECG Data Safety Analysis Set

| ECG parameter (unit)<br>Time point | dasiglucagon 0.3mg (N=XX) | dasiglucagon 0.6mg<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|
| ECG parameter (unit) | | | |
| Screening | | | |
| n | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |
| ••• | | | |
| Interpretation | | | |
| Screening | | | |
| Normal | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Abnormal (NCS) | XX ( XX.Xt) | 1111 ( 1111111111) | AA ( AA.AO) |

Percentages are based on the total number of patients in the safety analysis set.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

- 1) In general present mean to 1 decimal more than individual data, STD to 2 decimals more than individual data.
- 2) Order parameters as follows: Mean Heart Rate, PR Interval, QRS, QT, QTc, QTcF, and Interpretation.




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

Appendix C2: Study-Specific Shells for Section 16.2

16.2. Patient Data Listings

16.2.1 Discontinued Patients




Zealand Pharma A/S ZP4207-21052 Zealand Pharma A/S ZP4207-21052 Statistical Analysis Plan

2-Jan-25

Clinical Study Report
Page x of y

RUN DATE: DDMMMYYYY hh:mm

# Listing 16.2.1.1 Patient Disposition All Patients

| Treatment<br>Group | Patient<br>ID | Enrolled<br>Set <sup>[a]</sup> | Safety<br>Analysis<br>Set <sup>[b]</sup> | Full<br>Analysis<br>Set <sup>[c]</sup> | PK<br>Analysis<br>Set <sup>[d]</sup> | Date/Time at<br>Start of Dosing | Completed<br>Study | Completion or<br>Discontinuation<br>Date | Primary Reason for<br>Discontinuation from Study |
|---|---|---|---|---|---|---|---|---|---|
| Xxxx | xxxx | Yes/No | Yes/No | Yes/No | Yes/No | YYYY-MM-DDTHH:MM | Yes/No | YYYY-MM-DD | xxxxxxxx |

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Sort by Treatment group and Patient ID


<sup>[</sup>a] Requires parent's/legal guardian's agreement for the child to participate in a clinical trial following completion of the informed consent process and further that the child is screened and found eligible for the trial.

<sup>[</sup>b] All patients who were enrolled and received at least 1 dose of study drug.

<sup>[</sup>c] All patients of the safety analysis set.

<sup>[</sup>d] All patients with at least one quantifiable plasma concentration.


Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052
2-Jan-25

16.2.2 Protocol Deviations




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 Clinical Study Report Zealand Pharma A/S

Page x of y

RUN DATE: DDMMMYYYY hh:mm

2-Jan-25

# Listing 16.2.2.1 Protocol Deviations Safety Analysis Set

| | | Category for | | |
|---|---|---|---|---|
| Treatment | | Protocol | | |
| Group | Patient ID | Deviation | Protocol Deviation Coded Term | Protocol Deviation Term |
| xxxx | xxxx | xxxx | xxxx | xxxx |

This listing displays all study protocol deviations that are not COVID-19 related.

Source: xxx

ZP4207-21052

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Sort by Treatment group and Patient ID

2) Exclude COVID-19 related protocol deviations

3) SHELL ID: LPDEVV1




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 2-Jan-25 Clinical Study Report Zealand Pharma A/S ZP4207-21052

Page x of y

RUN DATE: DDMMMYYYY hh:mm

# Listing 16.2.2.2 COVID-19 Related Protocol Deviations Safety Analysis Set

| Treatment | | Category for<br>Protocol | | |
|---|---|---|---|---|
| Group | Patient ID | Deviation | Protocol Deviation Coded Term | Protocol Deviation Term |
| xxxx | xxxx | xxxx | xxxx | xxxx |

This listing displays all study protocol deviations that are COVID-19 related.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Sort by Treatment group and Patient ID

- 2) Include COVID-19 related protocol deviations only
- 3) SHELL ID: LPDEVV1




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 Clinical Study Report Zealand Pharma A/S

Page x of y

2-Jan-25

Listing 16.2.2.3 Patients not Fulfilling at least one Inclusion/Exclusion Criteria All Screened Patients

| Treatment | | | Inclusion/Exclusion | |
|---|---|---|---|---|
| Group | Patient ID | Date/Time of Informed Consent | Criterion Short Name | Inclusion/Exclusion Criterion |
| xxxx | xxxx | YYYY-MM-DD | INCL2 / EXCL3 | xxxxxxxxx |

Source: xxx

ZP4207-21052

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY RUN DATE: DDMMMYYYY hh:mm

Programming Note:

1) Sort by treatment group and patient




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052
2-Jan-25

16.2.3 Patients Excluded from the Analysis




 Zealand Pharma A/S
 Statistical Analysis Plan

 ZP4207-21052
 2-Jan-25

 Zealand Pharma A/S
 Clinical Study Report

Page x of y

# Listing 16.2.3.1 Patients Excluded from Analysis All Enrolled Patients

| | | | · | | | Excluded | |
|---|---|---|---|---|---|---|---|
| | | Excluded from | n. | Excluded from | | from PK | |
| Treatment | | Safety | Reason for Exclusion | Full Analysis | Reason for Exclusion | Analysis | Reason for Exclusion |
| Group | Patient ID | Analysis Set | from Safety Analysis Set | Set | from Full Analysis Set | Set | from PK Analysis Set |
| xxxx | xxxx | Yes/No | xxxxxxxxxxx | Yes/No | xxxxxxxxxxx | Yes/No | xxxxxxxxxxx |

Source: xxx

ZP4207-21052

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY hh:mm

Programming Note:

1) Sort by treatment group and patient




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

16.2.4 Demographic Data




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 2-Jan-25 Clinical Study Report Zealand Pharma A/S ZP4207-21052

Page x of y

RUN DATE: DDMMMYYYY hh:mm

# Listing 16.2.4.1 Demographic and Baseline Characteristics Safety Analysis Set

| Treatment<br>Group | Patient<br>ID | Re-screened<br>Patient?:<br>Previous<br>Patient ID | Date/Time<br>of Informed | Date of<br>Birth | Age<br>(years) | Sex | Ethnicity | Race | Date of<br>Diabetes<br>Diagnosis | Protocol<br>Version<br>Originally<br>Consented<br>to |
|---|---|---|---|---|---|---|---|---|---|---|
| хххх | xxxx | Y: XXXXX<br>N | YYYY-MM-DD | YYYY-MM-DD | xxx | Male/<br>Female/<br>Unknown/<br>Undifferentiated | Hispanic or Latino/<br>Not Hispanic or<br>Latino/<br>Not Reported/<br>Not Allowed to Ask<br>per Local<br>Regulation | xxxxx | YYYY-MM-D | D xxxxxxxxxx |

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Sort by treatment group and patient




Zealand Pharma A/S ZP4207-21052 Zealand Pharma A/S

ZP4207-21052

Statistical Analysis Plan
2-Jan-25
Clinical Study Report
Page x of y

RUN DATE: DDMMMYYYY hh:mm

# Listing 16.2.4.2 Medical History Safety Analysis Set

| Treatment | | Reported Term/ | Body System or System | Start Date of Medical | End Date of Medica | alEnd Relative to |
|---|---|---|---|---|---|---|
| Group | Patient ID | MedDRA Preferred Term | Organ Class | History Event | History Event | Reference Period |
| | | | | YYYY-MM-DD/ | YYYY-MM-DD/ | |
| xxxx | xxxx | xxxx | xxxx | Unknown | Unknown | ONGOING |

Terms are coded using MedDRA, version 24.1.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Sort by treatment group, patient and start date




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 Zealand Pharma A/S Clinical Study Report ZP4207-21052

Page x of y

RUN DATE: DDMMMYYYY hh:mm

2-Jan-25

## Listing 16.2.4.3 Prior and Concomitant Medications Safety Analysis Set

| Treatment<br>Group | Patient<br>ID | СМ# | P/<br>C | Medication<br>Name/<br>Preferred Name | Start Date<br>(Study Day) | End Date<br>(Study Day) | Dose<br>(unit) | Route of<br>Administration | Infusion<br>Rate<br>(mg/min) | Frequency | Indication<br>(Event ID/Specify) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xx | P/<br>C | xxxxx/<br>xxxxx | YYYY-MM-DD<br>(Day XX) | YYYY-MM-DD<br>(Day XX)<br>ONGOING | xxxx<br>(xx) | xxxxxx | xxx<br>NA | xxxx | Medical History (X)<br>Adverse Event (X)<br>Other (xxxxx) |

P: Prior medication C: Concomitant medication, #= number. Study day is derived relative to the date/time of start of study drug administration.

Terms are coded using WHODrug Global B3 format, Sep2021 release.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

Sort by treatment group, patient and CM#

2) Study day is derived relative to the date/time of start of study drug administration.




Zealand Pharma A/S

<u>ZP4207-21052</u>

Zealand Pharma A/S

zP4207-21052

2-Jan-25
Clinical Study Report
Page x of y

RUN DATE: DDMMMYYYY hh:mm

Statistical Analysis Plan

## Listing 16.2.4.4 Current Diabetes Treatment Safety Analysis Set

| Treatment | | Diabetes Medication/ | | | |
|---|---|---|---|---|---|
| Group | Patient ID | Preferred Name | Start Date (Study Day) | Dose (unit) | Route of Administration |
| | | xxxxx/ | | | |
| xxxx | xxxxx | xxxxx | YYYY-MM-DD (Day XX) | xxxx (xx) | xxxxxx |

Study day is derived relative to the date/time of start of study drug administration. Terms are coded using WHODrug Global B3 format, Sep2021 release.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

1) Sort by treatment group, patient and CM#

2) Study day is derived relative to the date/time of start of study drug administration.




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052
2-Jan-25

16.2.5 Compliance and/or Drug Concentration Data




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052

Clinical Study Report Zealand Pharma A/S Protocol Number: ZP4207-21052

2-Jan-25 Page x of y

RUN DATE: DDMMMYYYY hh:mm

# Listing 16.2.5.1 Study Drug Administration Safety Analysis Set

| | | Was | | Study Treatment<br>Label Identifier | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | | Dasiglucagon | Reason Not | (DUN)/ | Dosing | | | Route of | |
| Group | Patient ID | Admnistered? | Administered | Lot Number | Date/Time | Dose | (unit) | Administration | Location |
| xxxx | xxxxx | Yes/<br>No | xxxxxxxx | xxxxx/<br>xxxx | YYYY-MM-<br>DD/HH:MM | xxx | (xx) | Subcutaneous injection | Buttock<br>xxxxxxx |

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

1) Sort by treatment group and patient number




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052

Clinical Study Report Zealand Pharma A/S Protocol Number: ZP4207-21052

Page x of y

RUN DATE: DDMMMYYYY hh:mm

2-Jan-25

## Listing 16.2.5.2 Diabetes treatment prior hypoglycemia induction - MDI user Safety Analysis Set

| Treatment<br>Group | Patient ID | Date/ Time of last basal dose before the<br>Hypoglycemia procedure | Dose of last basal<br>dose<br>(IU) | Reduction of last basal dose<br>compared to the dose before<br>(%) |
|---|---|---|---|---|
| xxxx | xxxxx | YYYY-MM-DDTHH:MM | Xxxxx | Xxxxx |

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

1) Sort by treatment group and patient number




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
2-Jan-25

Zealand Pharma A/S
Protocol Number: ZP4207-21052
Page x of y

Listing 16.2.5.3 Diabetes treatment prior hypoglycemia induction - meal-time/ bolus insulins Safety Analysis Set

| Treatment<br>Group | Patient ID | Bolus Insulin name | Date/Time of bolus(es)<br>within 8 hours before<br>Hypoglycemia procedure | Dose of last bolus dose within 8 hours before Hypoglycemia procedure (enter 0 if none given): |
|---|---|---|---|---|
| xxxx | xxxx | Xxxx | YYYY-MM-DDTHH:MM | xxxx |

RUN DATE: DDMMMYYYY hh:mm

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

1) Sort by treatment group and patient number




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 2-Jan-25

Zealand Pharma A/S

Clinical Study Report Protocol Number: ZP4207-21052 Page x of y

## Listing 16.2.5.4 Diabetes treatment prior hypoglycemia induction - pump user Safety Analysis Set

| Treatment<br>Group | Patient ID | Insulin brand name | Date/Time of stopping<br>insulin pump before<br>initiation of<br>Hypoglycemia procedure | Total amount of insulin infused<br>6 hours before initiating<br>Hypoglycemia procedure<br>(IU) |
|---|---|---|---|---|
| xxxx | xxxxx | Xxxx | YYYY-MM-DDTHH:MM | xxxx |

RUN DATE: DDMMMYYYY hh:mm

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

1) Sort by treatment group and patient number




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052

Clinical Study Report Zealand Pharma A/S Protocol Number: ZP4207-21052

Page x of y

RUN DATE: DDMMMYYYY hh:mm

2-Jan-25

# Listing 16.2.5.5 Hypoglycemia Induction Procedure Safety Analysis Set

| | | | | Insulin | Infusion | | | Glucose Admi | nistration | ı |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Confirmatory | | | Plasma | Start | |
| | | | | Time | Plasma | | | Glucose | Time/ | |
| | | Time | Plasma Glucose | Insulin | Glucose | Total | Glucose | Before | Stop Time | Total |
| | | Procedure | Before Start | Infusion | Before | Insulin | Administered | Glucose | of | Glucose |
| Treatment | Patient | Was | of Procedure | Was | Dosing | Administered | Prior to | Infusion | Glucose | Administered |
| Group | ID | Initiated | (Unit) | Stopped | (Unit) | (IU) | Dosing? | (Unit) | Infusion | (mL) |
| xxxxx | xxxxx | HH:MM | | | xxxxx | xxx | Y/ | | HH:MM/ | |
| | | | xxxxxx (xxxx) | HH:MM | (xxxx) | | N | xxx (xxxx) | HH:MM | xxxxx |

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

2) Sort by treatment group and patient number




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
2-Jan-25

 ZP4207-21052
 2-Jan-25

 Zealand Pharma A/S
 Clinical Study Report

 Protocol Number: ZP4207-21052
 Page x of y

## Listing 16.2.5.6 dasiglucagon Plasma Concentrations Safety Analysis Set

| Treatment<br>Group | Patient<br>ID | Analyte (Unit) | Planned Timepoint | Not Done:<br>Reason | Date/Time of<br>Sample Collection | Elapsed Time<br>(Minutes) | Concentration |
|---|---|---|---|---|---|---|---|
| | | dasiglucagon | | | | | |
| XXXX | XXXX | (pmol/L) | Predose | | YYYY-MM-DDTHH: MM | -0.02 | XX.X |
| | | | 10 minutes post dose | Y: xxxxxxxx | | | |
| | | | 20 minutes post dose | | YYYY-MM-DDTHH:MM | 0.34 | XX.X |
| | | | 30 minutes post dose | | YYYY-MM-DDTHH:MM | 0.51 | XX.X |
| | | | 40 minutes post dose | | YYYY-MM-DDTHH:MM | 0.68 | XX.X |
| | | | 60 minutes post dose | | YYYY-MM-DDTHH:MM | 1.02 | XX.X |

RUN DATE: DDMMMYYYY hh:mm

dasiglucagon plasma concentrations at the Visit 2 (Dosing) visit. Concentration values are displayed to 3 significant figures.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

1) Sort by treatment group, patient number and planned timepoint.




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S

Clinical Study Report

Protocol Number: ZP4207-21052 Page x of y

## Listing 16.2.5.7 dasiglucagon PK Parameters Safety Analysis Set

| Treatment<br>Group | Patient ID | Parameter (unit) | Result | Status | Reason Not Done |
|---|---|---|---|---|---|
| xxxx | xxxx | T <sub>max</sub> (h) AUC <sub>0-20</sub> ( <unit>)</unit> | xxx | NOT DONE | xxxxx |
| | | | ••• | | • • • |

RUN DATE: DDMMMYYYY hh:mm

Results are displayed to 3 significant figures.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

1) Complete for each PK parameter listed in the SAP.

2) Sort by treatment group, patient and parameter (according to the order in section 12.1 of the SAP)>.




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052

Zealand Pharma A/S Protocol Number: ZP4207-21052 Clinical Study Report Page x of y

2-Jan-25

# Listing 16.2.5.8 Continuous Glucose Monitoring Safety Analysis Set

| Treatment<br>Group | Patient ID | Collection Date | Collection Time | Result | Unit |
|---|---|---|---|---|---|
| xxxx | xxxx | YYYY-MM-DD | HH:MM | xx.x | mg/dL |

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

Programming note:

1) Sort by treatment group, patient number, Visit, Date/ Time




 Zealand Pharma A/S
 Statistical Analysis Plan

 ZP4207-21052
 2-Jan-25

 Zealand Pharma A/S
 Clinical Study Report

Clinical Study Report
Page x of y

RUN DATE: DDMMMYYYY hh:mm

Listing 16.2.5.9 Glucose Analyzer data Safety Analysis Set

| Treatment<br>Group | Patient ID | Visit | Collection Date | Collection Time | Result | Unit |
|---|---|---|---|---|---|---|
| xxxx | xxxx | Dosing | YYYY- <b>MM</b> -DD | нн : мм | xx.x | xxx |
| | xxxx | | | | | |

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

Protocol Number: ZP4207-21052

1) Sort by treatment group, patient number, Date/time




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

16.2.6 Individual Efficacy Response Data




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
2-Jan-25

Zealand Pharma A/S

Clinical Study Report
Page x of y

RUN DATE: DDMMMYYYY hh:mm

Protocol Number: ZP4207-21052

#### Listing 16.2.6.1 Plasma Glucose Concentrations Safety Analysis Set

| | | | | | | | Change | |
|---|---|---|---|---|---|---|---|---|
| Treatment | | Parameter | | Date/Time of Collection | Plasma Glucose | Completion | from | Normal |
| Group | Patient ID | (unit) | Time Point[a] | (Study Day <sup>[b]</sup> ) | (mg/dL) [c] | Status | Baseline | Range |
| | | | | | | | xxxx or | |
| | | | | | | | -/xxxx <sup>[d]</sup> | |
| xxxx | xxxx | xxxx | Pre-dose (BL) | YYYY-MM-DDTHH:MM (Day XX) | xxxx (L) | | | xx-xx |
| | | | 10 min | YYYY-MM-DDTHH:MM (Day XX) | xxxx (H) | | | xx-xx |
| | | XXXX | Pre-dose | | | NOT DONE | | |

<sup>[</sup>a] BL: Baseline Flag

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Sort by treatment group, patient, then date/time.


<sup>(</sup>b) Study day is derived relative to the date/time of start of study drug administration.

<sup>[</sup>c] L: Below Normal Range, H: Above Normal Range

<sup>[</sup>d] Change to last recorded value prior to study drug administration / Change to recorded value at the nominal time point 'pre-dose' if different



Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

16.2.7 Adverse Event Listings




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S

Protocol Number: ZP4207-21052

Page x of y

#### Listing 16.2.7.1 Adverse Events Safety Analysis Set

| Treatment<br>Group - | | | System Organ | Start Date Time<br>(Study Day[b])/ | | | Action<br>Taken<br>with | | AESI <sup>[d]</sup> / | | | | | sma<br>cose |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>ID | | TE-<br>AE[a] | Preferred Term/ | End Date Time<br>(Study Day[b]) | SAE | Severity/<br>Causality | Study | Outcome | Important | Type of Other<br>Important Event <sup>[e]</sup> | | Start<br>Time | | Value<br>(unit) |
| XXXX | xx | Y/<br>N | xxxx/<br>xxxx/<br>xxxx | YYYY-MM-DDTHH:MM<br>(Day XX)/<br>YYYY-MM-DD-<br>DDTHH:MM<br>(Day XX) | Y | Mild/<br>Possible | Dose<br>Reduced | Unknown | N/<br>Y | Infection/ Overdose/ Abuse or misuse/ Error/ Accidental exposure/ Risk of liver injury | Y | HH:MM | xxxxx | (xxx) |
| | | | | YYYY-MM-DD<br>(Day XX)/<br>UNKNOWN | | | | | | | | | | |

#= number.

[a] TEAE: Treatment-emergent AE

[b] Study day is derived relative to the date/time of start of study drug administration.

[c] SAE: Serious AE

[d] AESI: AE of special interest

[e] Infection=Suspicion of transmission of infectious agents via the trial product; Overdose=Overdose of the trial product; Abuse or misuse=Suspected abuse or misuse of the trial product; Error=Medication error involving the trial product; Accidental exposure=Inadverdent or accidental exposure to the trial product; Risk of liver injury=Risk of liver injury defined as ALT or AST > 3 x ULN and total bilirubin > 2 x ULN, where no alternative etiology exists;

RUN DATE: DDMMMYYYY hh:mm

[f] Hypoglycemia Episode?

Adverse events were coded using MedDRA version 24.1.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

1) Sort by treatment group, patient, start date and end date.




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S

Page x of y

RUN DATE: DDMMMYYYY hh:mm

Zealand Pharma A/S
Protocol Number: ZP4207-21052

#### Listing 16.2.7.2 Adverse Events of Special Interest Safety Analysis Set

#= number.

- [a] TEAE: Treatment-emergent AE
- [b] Study day is derived relative to the date/time of start of study drug administration.
- [c] SAF. Serious AF
- [d] Infection=Suspicion of transmission of infectious agents via the trial product; Overdose=Overdose of the trial product; Abuse or misuse=Suspected abuse or misuse of the trial product; Error=Medication error involving the trial product; Accidental exposure=Inadverdent or accidental exposure to the trial product; Risk of liver injury=Risk of liver injury defined as ALT or AST > 3 x ULN and total bilirubin > 2 x ULN, where no alternative etiology exists;

[e] Hypoglycemia Episode?

Adverse events were coded using MedDRA version 24.1.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

- 1) Repeat Listing 16.2.7.1 for AESIs only
- 2) Remove AESI[d] variable
- 3) Update indexes [d] and [e] in column headers per footnotes above
- 4) Sort by treatment group, patient, start date and end date.




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052

Zealand Pharma A/S Clinical Study Report Protocol Number: ZP4207-21052

Page x of y

RUN DATE: DDMMMYYYY hh:mm

2-Jan-25

## Listing 16.2.7.3 Hemodynamic Changes During Adverse Events of Special Interest Safety Analysis Set

| | Start | | | | | | I I | <b>1</b> easur | rements Du | ring | The Event | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Date | | | | | | | H | ighest | 1 | Lowest | H | ighest | | Cowest |
| | Time | | | Hig | hest | L | owest | Sys | tolic BP | Sys | tolic BP | Dia | astolic | Di | astolic |
| | (Study | 7 | | Pulse | (bpm) | Puls | e (bpm) | ( | (mmHg) | | (mmHg) | BP | (mmHg) | BP | (mmHg) |
| | Day[a]) | / Event | | | | | | | | | | | | | |
| | End Da | ate Associate | d | | | | | | | | | | | | |
| | (Study | y With Any | | | | | | | | | | | | | |
| Treatment Group - | · Day[a]) | Signs Or | | | | | | | | | | | | | |
| Patient ID | AE# | Symptoms? | Narrative | <b>Value</b> D | ate/Time | Value: | Date/Time | Value | eDate/Time | Value | eDate/Time | Value | Date/Time | Value | Date/Tim |
| xxxx | xx YYYY-1 | MM-Y: | xxxxxxxx | XX Y | YYY-MM- | xx | YYYY-MM- | xxx | YYYY-MM- | xxx | YYYY-MM- | xxx | YYYY-MM- | xxx | YYYY-MM- |
| | DDTHH | : MM xxxxxxxx | | | DD/ | | DD/ | | DD/ | | DD/ | | DD/ | | DD/ |
| | (Day | | | | HH:MM | | HH:MM | | HH:MM | | HH:MM | | HH:MM | | HH:MM |
| | XX)/ | | | | | | | | | | | | | | |
| | YYYY-1 | -MM | | | | | | | | | | | | | |
| | DD | | | | | | | | | | | | | | |
| | (Day 1 | XX) | | | | | | | | | | | | | |
| | | N | | | | | | | | | | | | | |

#= number.

[a] Study day is derived relative to the date/time of start of study drug administration.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

Sort by treatment group, patient and AE#.




 Zealand Pharma A/S
 Statistical Analysis Plan

 ZP4207-21052
 2-Jan-25

 Zealand Pharma A/S
 Clinical Study Report

Zealand Pharma A/S Clini Protocol Number: ZP4207-21052

Page x of y

RUN DATE: DDMMMYYYY hh:mm

#### Listing 16.2.7.4 Other Important Events Safety Analysis Set

#= number.

- [a] TEAE: Treatment-emergent AE
- [b] Study day is derived relative to the date/time of start of study drug administration.
- [c] SAE: Serious AF
- [d] Infection=Suspicion of transmission of infectious agents via the trial product; Overdose=Overdose of the trial product; Abuse or misuse=Suspected abuse or misuse of the trial product; Error=Medication error involving the trial product; Accidental exposure=Inadverdent or accidental exposure to the trial product; Risk of liver injury=Risk of liver injury defined as ALT or AST > 3 x ULN and total bilirubin > 2 x ULN, where no alternative etiology exists;

[e] Hypoglycemia Episode?

Adverse events were coded using MedDRA version 24.1.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

- 1) Repeat Listing 16.2.7.1 for Other Important Events only
- 2) Remove Other Important Event? variable
- 3) Sort by treatment group, patient, start date and end date.




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S

Protocol Number: ZP4207-21052 Page x of y

## Listing 16.2.7.5 Details of Other Important Events Safety Analysis Set

| Treatment<br>Group | Patient ID | Other Important Event | Description of Event | Start Date Time<br>(Study Day[a])/ | End Date<br>(Study Day <sup>[a]</sup> ) | Event Related to an AE or SAE [b]? |
|---|---|---|---|---|---|---|
| xxxx | xxxx | Suspicion of transmission of<br>infectious agents via the<br>trial product | ****** | YYYY-MM-DDTHH:MM<br>(Day XX) | YYYY-MM-DDTHH:MM<br>(Day XX) | Y/N |

RUN DATE: DDMMMYYYY hh:mm

[a] Study day is derived relative to the date/time of start of study drug administration.

[b] SAE: Serious AE

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

1) Sort by treatment group, patient, start date and end date.




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052
2-Jan-25

Zealand Pharma A/S
Protocol Number: ZP4207-21052

Clinical Study Report
Page x of y

## Listing 16.2.7.6 Local Tolerability Assessment Safety Analysis Set

| | | | Date of | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Assessmen | | Were any | | | Reaction | | | | Likely |
| 'reatmer | nt Patien | t | (Study | Planned | reactions | Time of | Type of | Observed at | | | Action | Cause of |
| Group | ID | Visit | Day <sup>[a]</sup> ) | Timepoint | observed? | Assessment | Reaction | Injection Sit | e? Severit | y AE | † Taken | Reaction |
| | | | YYYY-MM-D | D | | | | | | | | |
| | | | (Day XX) | 30 minutes | 5 | | Spontaneous | | | | | |
| xxx | xxxx | Dosing | | post-dose | Y | HH:MM | Pain | N | | | | |
| | | | | | | | | | | | Other: | Insertion |
| | | | | | | HH:MM | Other: xxxxxx | Y | Mild | xx | xxxx | Site |
| | | Follow-up | | | | | | | | | | |
| | | | | | Y | | Spontaneous | | | | No Action | |
| | | | | | | HH:MM | Pain | Y | Severe | xx | Taken | Drug |
| | | | | 30 minutes | | | | | | | | |
| | | Dosing | | post-dose | N | | | | | | | |

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

Programming note:

1) Sort by treatment group, patient, date, planned timepoint, time and type of reaction.


<sup>[</sup>a] Study day is derived relative to the date/time of start of study drug administration.



Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S

Clinical Study Report

Zealand Pharma A/S
Protocol Number: ZP4207-21052
Page x of y

## Listing 16.2.7.7 Death Details Safety Analysis Set

Treatment

RUN DATE: DDMMMYYYY hh:mm

[a] Study day is derived relative to the date/time of start of study drug administration.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note:

1) Sort by treatment group and patient.




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 2-Jan-25 Page x of y

Protocol Number: ZP4207-21052

# Listing 16.2.7.8 Adverse Events for Screening Failures Screening Failures

Programming note:

1) Repeat Listing 16.2.7.1 for AEs for screening failures (i.e. not belonging to the safety set)




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

16.2.8 Listing of Individual Laboratory Measurements by Subject, When Required by Regulatory Authorities




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
2-Jan-25

Zealand Pharma A/S

Protocol Number: ZP4207-21052

Clinical Study Report Page x of y

RUN DATE: DDMMMYYYY hh:mm

## Listing 16.2.8.1 Hematology Safety Analysis Set

| Treatment<br>Group | Patient ID | Parameter<br>(unit) | Visit <sup>[a]</sup> | Date/Time of Collection (Study Day <sup>[b]</sup> ) | Result <sup>[c]</sup> | Completion<br>Status | Change<br>from<br>Baseline | Normal<br>Range |
|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx | xxxx | Screening (BL) | YYYY-MM-DDTHH:MM (Day XX) | xxxx (L) | | xxxx | xx-xx |
| | | | Follow-up | YYYY-MM-DDTHH:MM (Day XX) | xxxx (H) | | | xx-xx |
| | | xxxx | Screening | | | NOT DONE | | |

[a] BL: Baseline Flag

[c] L: Below Normal Range, H: Above Normal Range

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Sort by treatment group, patient, then Laboratory parameter (alphabetically), then date/time.

2) After each parameter, add a blank line


<sup>[</sup>b] Study day is derived relative to the date/time of start of study drug administration.



Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S

Protocol Number: ZP4207-21052 Page x of y

## Listing 16.2.8.2 Chemistry Safety Analysis Set

RUN DATE: DDMMMYYYY hh:mm

[a] BL: Baseline Flag

[b] Study day is derived relative to the date/time of start of study drug administration.

[c] L: Below Normal Range, H: Above Normal Range

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Repeat Listing 16.2.8.1 for Chemistry parameters.

- 2) Sort by treatment group, patient, then Laboratory parameter (alphabetically), then date/time.
- 3) After each parameter, add a blank line
- 4) Plasma glucose concentrations should be included in Listing 16.2.6.1 only




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S

Protocol Number: ZP4207-21052 Page x of y

## Listing 16.2.8.3 Coagulation Safety Analysis Set

RUN DATE: DDMMMYYYY hh:mm

[a] BL: Baseline Flag

[b] Study day is derived relative to the date/time of start of study drug administration.

[c] L: Below Normal Range, H: Above Normal Range

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming Note:

1) Repeat Listing 16.2.8.1 for Coagulation.

- 2) Sort by treatment group, patient, then Laboratory parameter (alphabetically), then date/time.
- 3) After each parameter, add a blank line




Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
ZP4207-21052

16.2.9 Other Data




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 2-Jan-25

Clinical Study Report Zealand Pharma A/S Protocol Number: ZP4207-21052

Page x of y

## Listing 16.2.9.1 Vital Signs Safety Analysis Set

| Treatmen | t Patient | Parameter | | | Date Time of Asse | ssment | Completion | | Change<br>from | |
|---|---|---|---|---|---|---|---|---|---|---|
| Group | ID | (unit) | Visit[a] | Time Point | (Study Day[b]) | | Status | Result | Baseline | Location |
| xxxx | xxxx | xxxx | Screening | | YYYY-MM-DDTHH:MM | (Day XX) | | xxxx | xxxx | Axilla |
| | | | Dosing (BL) | Pre dose | $\verb"YYYY-MM-DDTHH:MM"$ | (Day XX) | | | | Rectum |
| | | | | 30 minutes post-dose | | | Not Done | | | |
| | xxxx | <br>Interpretation | <br>Screening | | YYYY-MM-DDTHH:MM | (Day XX) | | Abnormal | | |
| | | | Dosing (BL) | Pre dose | YYYY-MM-DDTHH:MM | (Day XX) | | Abnormal<br>(NCS) | | |
| | | • • • | | • • • • | ••• | | | • • • • | | |

<sup>[</sup>a] BL: Baseline Flag

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

#### Programming Note:

- 1) Sort by treatment group, patient, then parameter (Height, Weight, BMI, Temperature, Systolic BP, Diastolic BP, Pulse, Interpretation), then date/time.
- 2) After each parameter, add a blank line


<sup>[</sup>b] Study day is derived relative to the date/time of start of study drug administration.



Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052

Zealand Pharma A/S Clinical Study Report

Protocol Number: ZP4207-21052 Page x of y

## Listing 16.2.9.2 Physical Examination Safety Analysis Set

| Treatment<br>Group | Patient ID | Body System | Visit <sup>[a]</sup> | Date Time of Exam (Study Day [b]) | Completion Status | Result |
|---|---|---|---|---|---|---|
| xxxx | xxxx | HEAD, EARS, EYES, NOSE,<br>THROAT INCLUDING THYROID<br>GLAND | Screening (BL) | YYYY-MM-DDTHH:MM (Day XX) | | Normal |
| | | | Dosing | YYYY-MM-DDTHH:MM (Day XX) | | Abnormal (CS) |
| | | | Follow-up | | Not Done | |
| | xxxx | ALL PHYSICAL EXAMINATIONS | Screening | | Not Done | ••• |

<sup>[</sup>a] BL: Baseline Flag

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

2-Jan-25

#### Programming Note:

- 1) Sort by treatment group, patient, then parameter (match the order in the CRF), then date/time.
- 2) After each parameter, add a blank line


<sup>[</sup>b] Study day is derived relative to the date/time of start of study drug administration.



Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052

Zealand Pharma A/S Protocol Number: ZP4207-21052

Clinical Study Report Page x of y

2-Jan-25

## Listing 16.2.9.3 Electrocardiogram Safety Analysis Set

| Treatment Patient Parameter | | | | Date Time of Assessment | Completion | Reason Not | : | Specify<br>Abnormal | |
|---|---|---|---|---|---|---|---|---|---|
| Group | ID | (unit) | Visit | (Study Day <sup>[a]</sup> ) | Position | Status | Done | Result | Findings |
| xxxx | xxxx | xxxx | Screening | YYYY-MM-DDTHH:MM (Day XX) | Supine | | | xxxx | |
| | | <br>Interpretation | <br>n | | ••• | | | <br>Abnormal (CS) | xxxxxxxx |
| | xxxx | ALL ECG TESTS | <br>Screening | | | Not Done | xxxxxxx | | |
| | | ••• | | | | | | ••• | |

<sup>[</sup>a] Study day is derived relative to the date/time of start of study drug administration.

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

RUN DATE: DDMMMYYYY hh:mm

#### Programming Note:

- 1) Sort by treatment group, patient, then parameter (Heart Rate, PR Interval, QRS, QT, QTcF, and Interpretation) then date/time.
- 2) After each patient, add a blank line




Zealand Pharma A/S

ZP4207-21052
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S
Zealand Pharma A/S

Clinical Study Report
Page x of y

Protocol Number: ZP4207-21052

Listing 16.2.9.4 Hospitalization
Safety Analysis Set

Treatment

Group Patient ID Date of Admission (Study Day[a]) Date of Discharge (Study Day[a])

XXXX

[a] Study day is derived relative to the date/time of start of study drug administration.

YYYY-MM-DD (Day XX)

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY hh:mm

YYYY-MM-DD (Day XX)

Programming note: Sort by treatment group and patient.




Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052 2-Jan-25 Clinical Study Report

Zealand Pharma A/S Protocol Number: ZP4207-21052

## Listing 16.2.9.5 Immunogenicity Safety Analysis Set

Page x of y

RUN DATE: DDMMMYYYY hh:mm

| Treatment | Patient | | | Date Time of Assessment | Completion | Reason Not | |
|---|---|---|---|---|---|---|---|
| Group | ID | Parameter (unit) | Visit <sup>[a]</sup> | (Study Day <sup>[b]</sup> ) | Status | Done | Result |
| | | | | | | | xxxx |
| xxxx | xxxx | xxxx | Screening (BL) | YYYY-MM-DDTHH:MM (Day XX) | | | xxxx |
| | | | Follow-up | YYYY-MM-DDTHH:MM (Day XX) | | | xxxx |
| | <br>xxxx | <br>All Immunogenicity<br>Tests | <br>7<br>xxxx | | Not Done | xxxxxxx | |

<sup>[</sup>a] BL: Baseline Flag

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY

Programming note: Sort by treatment group, patient, parameter and visit.


<sup>[</sup>b] Study day is derived relative to the date/time of start of study drug administration.



Zealand Pharma A/S Statistical Analysis Plan ZP4207-21052

Zealand Pharma A/S

Clinical Study Report Page x of y

2-Jan-25

Protocol Number: ZP4207-21052

# Listing 16.2.9.6 Food and Drink Intake Safety Analysis Set

| | | | | Pre Dose | Post Dose | | |
|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Patient<br>ID | Visit | Did Patient Refrain from Food/Drink <sup>[a]</sup> ? Reason If No | Date | Time of Last Food/Drink[b] | Did Patient Take Any<br>Food/Drink During Follow-<br>up? | Time of Food/Drink(b) |
| xxx | xxxx | Dosing | Y | YYYY-MM-DD | HH:MM | N | |
| | xxxx | Dosing | N: xxxxxxx | YYYY-MM-DD | HH:MM | Y | HH:MM,<br>HH:MM,<br>HH:MM, |

<sup>[</sup>a] Except water, for 4 hours prior to dosing

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY RUN DATE: DDMMMYYYY hh:mm

Programming note: Sort by treatment group and patient. Add a blank line between patients.


<sup>[</sup>b] Excluding water



Zealand Pharma A/S
ZP4207-21052
Statistical Analysis Plan
2-Jan-25

Zealand Pharma A/S

Protocol Number: ZP4207-21052

Clinical Study Report
Page x of y

## Listing 16.2.9.7 Technical Complaints Safety Analysis Set

| Treatment<br>Group | Patient<br>ID | Date Technical<br>Complaint<br>Detected | Date<br>Technical<br>Complaint<br>Reported | Difficulties<br>Administering<br>Drug?: Details | Trial DUN Number | Action<br>Taken | Related to AE?: ID Yes: XX |
|---|---|---|---|---|---|---|---|
| xxxx | xxx | YYYY-MM-DD<br>YYYY-MM-DD | YYYY- <b>MM</b> -DD | Yes: Drug jammed | ***** | ***** | |
| | | IIII-MM-DD | YYYY- <b>MM</b> -DD | Yes: xxxxxxxxx | xxxxxxxx | xxxxxx | No |

Source: xxx

PROGRAM SOURCE: xxx.sas, DATA CUT-OFF DATE: DDMMMYYYY RUN DATE: DDMMMYYYY hh:mm

Programming note: Sort by treatment group, patient and date technical complaint detected
